CLINICAL TRIAL: NCT01072175
Title: An Open-Label, Dose-Escalation, Phase I/II Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Clinical Activity of the BRAF Inhibitor GSK2118436 in Combination With the MEK Inhibitor GSK1120212 in Subjects With BRAF Mutant Metastatic Melanoma
Brief Title: Investigate Safety, Pharmacokinetics and Pharmacodynamics of GSK2118436 & GSK1120212
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 113220
Record Dates: First submitted 2010-02-12; First posted 2010-02-19 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Cancer
Keywords: drug-drug interaction; BRAF inhibitor; expansion cohorts; melanoma; dose escalation; MEK inhibitor
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm Part A (Experimental): Day 1: GSK2118436 75mg; Day 2 through Day 16: GSK1120212 2mg; Day 15: GSK2118436 75mg +GSK1120212 2mg Drug-drug interaction
  Interventions: Drug: GSK2118436; Drug: GSK1120212
- Arm Part B (Experimental): GSK2118436 + GSK1120212 Dose escalation to a maximum tolerated combination dose
  Interventions: Drug: GSK2118436
- Arm Part C (Experimental): GSK2118436 + GSK1120212 cohort expansion for safety and efficacy
  Interventions: Drug: GSK2118436; Drug: GSK1120212

INTERVENTIONS:
Drug: GSK2118436 — GSK2118436 is a potent and selective inhibitor of BRAF kinase activity with a mode of action consistent with adenosine triphosphate-competitive inhibition.
Drug: GSK1120212 — GSK1120212 is a potent and highly selective inhibitor of MEK1/2 activation and kinase activity.
  Arms: Arm Part A; Arm Part C

SUMMARY:
This was an open-label, dose escalation study to investigate the safety, pharmacokinetics, pharmacodynamics and clinical activity of GSK2118436 and GSK1120212 in combination. This study was designed in four parts. In Part A, the effect of repeat doses of GSK1120212 on the pharmacokinetics of single dose GSK2118436 was investigated prior to evaluating combination regimens. In Part B, the range of tolerated dose combinations was identified using a dose-escalation procedure. In Part C, different dose combinations of GSK2118436 and GSK1120212 were evaluated, based on results from the dose escalation cohorts. In Part D, the pharmacokinetics and safety of GSK2118436 administered as HPMC capsules alone and in combination with GSK1120212 was evaluated.

DETAILED DESCRIPTION:
During Part A, a cohort of subjects received a single dose of GSK2118436 alone (Day 1) and then repeat doses of GSK1120212 for (Day 2 through Day 15). The dose regimen of GSK1120212 were continuous dosing. A second single dose of GSK2118436 was administered on Day 15 concomitantly with GSK1120212. Day 16 through Day 28 was a washout period, during which no study medication was administered. Starting on Day 29, subjects who elected to continue participation in the study were doses with GSK2118436. The dose of GSK2118436 after Day 29 might be altered based on emerging data from the first-time-in human study BRF112680. The dose might be increased to a dose level that has been completed and determined to be less than or equal to the maximum tolerated dose in that study.

Part B of the study enrolled cohorts in escalating doses to identify a set of allowable doses to be expanded in Part C. Subjects were enrolled in a 3+3 cohort design, with provisional dose levels of both drugs. The decision regarding escalation to the next dose levels of GSK1120212 and GSK2118436 was further guided by a Bayesian logistic regression model. The first cohort started at low doses for both drugs. Doses up to 300 mg/day for GSK2118436 and up to 3 mg QD for GSK1120212 were studied. The starting dose might be lowered based on emerging data from other studies and from Part A.

Expansion cohorts enrolled in Part C at dose levels of GSK2118436 and GSK1120212 as defined in Part B. One of the selected doses might include GSK2118436 administered as monotherapy at a tolerable dose (less than or equal to the maximum tolerated dose) determined in BRF112680. Part C was a randomized open-label Phase II portion of the study, and consisted of expansion cohorts investigating 2 to 3 dose levels of GSK2118436 and GSK1120212 dosing in combination, and GSK2118436 administered as monotherapy. Subjects were assigned to treatment arms in a randomized fashion to compare tolerability and safety. Population PK parameters, clinical activity, durability of response and safety of GSK2118436 and GSK1120212 dosed orally in combination and GSK2118436 as monotherapy were evaluated.

Part D consisted of evaluation of the pharmacokinetics of GSK2118436 HPMC capsules administered as monotherapy and in combination with GSK1120212. Pharmacokinetics of GSK2118436 was assessed following a single dose on Day 1 and after repeat dosing (Day 21) and compared between combination and monotherapy. The pharmacokinetics of GSK1120212 was also be assessed. Safety, tolerability and clinical activity were evaluated in 4 dosing cohorts. These cohorts might be expanded for additional safety data. Subjects were randomized to different cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Capable of given written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female age 18 years or greater; able to swallow and retain oral medication.
* BRAF mutation positive melanoma or colorectal cancer; other BRAF mutation positive tumor types may be considered.
* Measurable disease according to RECIST version 1.1.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1 for Parts A and B. Subjects with Eastern Cooperative Oncology Group Performance Status of 2 or less may be entered into Part C with approval of medical monitor.
* Agree to contraception requirements.
* Calcium phosphorus product less than 4.0mmol2/L2.
* Adequate organ system function.

Key Exclusion Criteria:

* Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy).
* Part A and Part B: Prior exposure to BRAF or MEK inhibitors unless approved by the GSK Medical Monitor.
* Part C: Prior exposure to BRAF or MEK inhibitors. Prior anti-cancer therapy in the metastatic setting, with the exception of up to one regimen of chemotherapy and/or interleukin-2 (IL-2).
* Part D: Prior exposure to BRAF inhibitors. A washout period of 6 weeks is required for ipilimumab.
* Received an investigational anti-cancer drug within 4 weeks or 5 half-lives (whichever is shorter) of study drug administration--- at least 14 days must have passed between the last dose of prior investigational anti-cancer drug and the first dose of study drug.
* Current use of a prohibited medication or requires any of these medications during treatment with study drug.
* Current use of therapeutic warfarin.
* Any major surgery, radiotherapy, or immunotherapy within the last 4 weeks. Limited radiotherapy within the last 2 weeks.
* Chemotherapy regimens with delayed toxicity within the last 4 weeks. Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.
* Unresolved toxicity greater than National Cancer Institute-Common Terminology Criteria for Adverse Events version 4 Grade 1 from previous anti-cancer therapy except alopecia.
* History of retinal vein occlusion, central serous retinopathy or glaucoma.
* Predisposing factors to retinal vein occlusion including uncontrolled hypertension, uncontrolled diabetes, uncontrolled hyperlipidemia, and coagulopathy.
* Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for retinal vein occlusion or central serous retinopathy.
* Intraocular pressure greater than 21mm Hg as measured by tonography.
* Glaucoma diagnosed within one month prior to study Day 1.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism or excretion of drugs.
* Known human immunodeficiency virus, Hepatitis B or Hepatitis C infection.
* Primary malignancy of the central nervous system.
* Untreated or symptomatic brain metastasis, leptomeningeal disease or spinal cord compression. Subjects who are on a stable dose of corticosteroids for more than 1 month or off corticosteroids for 2 weeks can be enrolled with approval of medical monitor. Subjects are not permitted to receive enzyme-inducing anti-epileptic drugs.
* Subjects with brain metastases are excluded, unless

  a. All known lesions must be previously treated with surgery or stereotactic radiosurgery, and- b. Brain lesion(s), if still present, must be confirmed stable (i.e. no increase in lesion size) for ≥90 days prior to first dose on study (must be documented with two consecutive MRI or CT scans using contrast), and c. Asymptomatic with no corticosteroids requirement for ≥ 30 days prior to first dose on study, and d. No enzyme-inducing anticonvulsants for ≥ 30 days prior to first dose on study.
* History of alcohol or drug abuse within 6 months prior to screening.
* Psychological, familial, sociological or geographical conditions that do not permit compliance with the protocol.
* QTc interval greater than or equal to 480msecs.
* History of acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting within the past 24 weeks.
* Class II, III, or IV heart failure as defined by the New York Heart Association functional classification system.
* Abnormal cardiac valve morphology (subjects with minimal abnormalities can be entered on study with approval from the medical monitor.
* Treatment refractory hypertension defined as a blood pressure of systolic> 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy
* Patients with intra-cardiac defibrillators or permanent pacemakers.
* Cardiac metastases
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study drugs or excipients.
* Pregnant or lactating female.
* Unwillingness or inability to follow the procedures required in the protocol.
* Uncontrolled diabetes, hypertension or other medical conditions that may interfere with assessment of toxicity.
* Subjects with known glucose 6 phosphate dehydrogenase deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2010-03-26 (Actual); Primary Completion 2012-05-31 (Actual); Study Completion 2018-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (11):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Lutherville-Timonium, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Flaherty KT, Infante JR, Daud A, Gonzalez R, Kefford RF, Sosman J, Hamid O, Schuchter L, Cebon J, Ibrahim N, Kudchadkar R, Burris HA 3rd, Falchook G, Algazi A, Lewis K, Long GV, Puzanov I, Lebowitz P, Singh A, Little S, Sun P, Allred A, Ouellet D, Kim KB, Patel K, Weber J. Combined BRAF and MEK inhibition in melanoma with BRAF V600 mutations. N Engl J Med. 2012 Nov 1;367(18):1694-703. doi: 10.1056/NEJMoa1210093. Epub 2012 Sep 29. PMID 23020132
- [Derived] Long GV, Eroglu Z, Infante J, Patel S, Daud A, Johnson DB, Gonzalez R, Kefford R, Hamid O, Schuchter L, Cebon J, Sharfman W, McWilliams R, Sznol M, Redhu S, Gasal E, Mookerjee B, Weber J, Flaherty KT. Long-Term Outcomes in Patients With BRAF V600-Mutant Metastatic Melanoma Who Received Dabrafenib Combined With Trametinib. J Clin Oncol. 2018 Mar 1;36(7):667-673. doi: 10.1200/JCO.2017.74.1025. Epub 2017 Oct 9. PMID 28991513
- [Derived] Long GV, Grob JJ, Nathan P, Ribas A, Robert C, Schadendorf D, Lane SR, Mak C, Legenne P, Flaherty KT, Davies MA. Factors predictive of response, disease progression, and overall survival after dabrafenib and trametinib combination treatment: a pooled analysis of individual patient data from randomised trials. Lancet Oncol. 2016 Dec;17(12):1743-1754. doi: 10.1016/S1470-2045(16)30578-2. Epub 2016 Nov 16. PMID 27864013
- [Derived] Long GV, Weber JS, Infante JR, Kim KB, Daud A, Gonzalez R, Sosman JA, Hamid O, Schuchter L, Cebon J, Kefford RF, Lawrence D, Kudchadkar R, Burris HA 3rd, Falchook GS, Algazi A, Lewis K, Puzanov I, Ibrahim N, Sun P, Cunningham E, Kline AS, Del Buono H, McDowell DO, Patel K, Flaherty KT. Overall Survival and Durable Responses in Patients With BRAF V600-Mutant Metastatic Melanoma Receiving Dabrafenib Combined With Trametinib. J Clin Oncol. 2016 Mar 10;34(8):871-8. doi: 10.1200/JCO.2015.62.9345. Epub 2016 Jan 25. PMID 26811525
- [Derived] Corcoran RB, Atreya CE, Falchook GS, Kwak EL, Ryan DP, Bendell JC, Hamid O, Messersmith WA, Daud A, Kurzrock R, Pierobon M, Sun P, Cunningham E, Little S, Orford K, Motwani M, Bai Y, Patel K, Venook AP, Kopetz S. Combined BRAF and MEK Inhibition With Dabrafenib and Trametinib in BRAF V600-Mutant Colorectal Cancer. J Clin Oncol. 2015 Dec 1;33(34):4023-31. doi: 10.1200/JCO.2015.63.2471. Epub 2015 Sep 21. PMID 26392102
- [Derived] Latimer NR, Amonkar MM, Stapelkamp C, Sun P. Adjusting for confounding effects of treatment switching in a randomized phase II study of dabrafenib plus trametinib in BRAF V600+ metastatic melanoma. Melanoma Res. 2015 Dec;25(6):528-36. doi: 10.1097/CMR.0000000000000193. PMID 26340744
- [Derived] Johnson DB, Flaherty KT, Weber JS, Infante JR, Kim KB, Kefford RF, Hamid O, Schuchter L, Cebon J, Sharfman WH, McWilliams RR, Sznol M, Lawrence DP, Gibney GT, Burris HA 3rd, Falchook GS, Algazi A, Lewis K, Long GV, Patel K, Ibrahim N, Sun P, Little S, Cunningham E, Sosman JA, Daud A, Gonzalez R. Combined BRAF (Dabrafenib) and MEK inhibition (Trametinib) in patients with BRAFV600-mutant melanoma experiencing progression with single-agent BRAF inhibitor. J Clin Oncol. 2014 Nov 20;32(33):3697-704. doi: 10.1200/JCO.2014.57.3535. Epub 2014 Oct 6. PMID 25287827
- [Derived] Frederick DT, Salas Fragomeni RA, Schalck A, Ferreiro-Neira I, Hoff T, Cooper ZA, Haq R, Panka DJ, Kwong LN, Davies MA, Cusack JC, Flaherty KT, Fisher DE, Mier JW, Wargo JA, Sullivan RJ. Clinical profiling of BCL-2 family members in the setting of BRAF inhibition offers a rationale for targeting de novo resistance using BH3 mimetics. PLoS One. 2014 Jul 1;9(7):e101286. doi: 10.1371/journal.pone.0101286. eCollection 2014. PMID 24983357
- [Derived] Carlino MS, Gowrishankar K, Saunders CA, Pupo GM, Snoyman S, Zhang XD, Saw R, Becker TM, Kefford RF, Long GV, Rizos H. Antiproliferative effects of continued mitogen-activated protein kinase pathway inhibition following acquired resistance to BRAF and/or MEK inhibition in melanoma. Mol Cancer Ther. 2013 Jul;12(7):1332-42. doi: 10.1158/1535-7163.MCT-13-0011. Epub 2013 May 3. PMID 23645591

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 16 sites: Australia (2) and USA (14)
Pre-assignment Details: The study was comprised of Parts A, B, and D, which constitute the Phase I part of the study, and Part C, which constitutes the randomized Phase II part of the study. Participants did not enroll in all parts of the study sequentially. Each part of the study was comprised of a separate population of participants.
Groups:
- Part A: Dabrafenib 75 mg + Trametinib 2 mg: Participants received a single dose of dabrafenib 75 mg gelatin capsules with repeat dose trametinib (Day 15).
- Part B: Dabrafenib 75 mg + Trametinib 1 mg: Melanoma BRAF-positive participants who did not receive prior treatment with BRAF inhibitors received dabrafenib 75 mg gelatin capsules BID and trametinib 1 mg tablets QD as continuous daily dosing. Dose escalation decisions were made based on all available pharmacokinetic (PK), safety, and other data from the first 4 evaluable participants, and additional participants were enrolled based on dose-limiting toxicities (DLTs) occurring during the first 3 weeks of treatment.
- Part B: Dabrafenib 150 mg + Trametinib 1 mg: Melanoma BRAF-positive participants who did not receive prior treatment with BRAF inhibitors and participants who had salivary ductal cancer received dabrafenib 150 mg gelatin capsules BID and trametinib 1 mg tablets QD as continuous daily dosing. Dose escalation decisions were made based on all available PK, safety, and other data from the first 4 evaluable participants and additional participants were enrolled based on DLTs occurring during the first 3 weeks of treatment.
- Part B: Dabrafenib 150 mg + Trametinib 1.5 mg: Melanoma BRAF-positive participants who did not receive prior treatment with BRAF inhibitors received dabrafenib 150 mg gelatin capsules BID and trametinib 1.5 mg tablets QD as continuous daily dosing. Dose escalation decisions were made based on all available PK, safety, and other data from the first 4 evaluable participants, and additional participants were enrolled based on DLTs occurring during the first 3 weeks of treatment.
- Part B: Dabrafenib 150 mg + Trametinib 2 mg: Melanoma BRAF-positive participants who received prior treatment with BRAF inhibitors and participants who had colorectal cancer and BRAFi naïve melanoma received dabrafenib 150 mg gelatin capsules BID and trametinib 2 mg tablets QD as continuous daily dosing. Dose escalation did not proceed beyond these doses of dabrafenib and trametinib.
- Part C (Randomized): Dabrafenib 150 mg: Participants received dabrafenib 150 mg gelatin capsules BID.
- Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg: Participants received dabrafenib 150 mg gelatin capsules BID and trametinib 1 mg tablets QD.
- Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg: Participants received dabrafenib 150 mg gelatin capsules BID and trametinib 2 mg tablets QD.
- Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg: Participants who received dabrafenib 150 mg capsules BID alone in the Randomized Phase were given the opportunity to receive combination dosing of dabrafenib 150 mg gelatin capsules BID and trametinib 2 mg tablets QD upon disease progression with approval of the GlaxoSmithKline (GSK) Medical Monitor.
- Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg: Participants received dabrefinib 75 mg HPMC capsules BID. These participants, after completion of serial PK collection in the first treatment period, were allowed to continue with dabrafenib 75 mg BID and trametinib 2 mg tablets QD as combination dosing starting on Day 29.
- Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg: Participants received dabrefinib 150 mg HPMC capsules BID. These participants, after completion of serial PK collection in the first treatment period, were allowed to continue with dabrafenib 150 mg BID and trametinib 2 mg tablets QD as combination dosing starting on Day 29.
- Part D: Dabrafenib 75 mg + Trametinib 2 mg: Participants received dabrefinib 75 mg HPMC capsules BID and trametinib 2 mg tablets QD.
- Part D: Dabrafenib 150 mg + Trametinib 2 mg: Participants received dabrefinib 150 mg HPMC capsules BID and trametinib 2 mg tablets QD.
Period: Part A (Drug-Drug Interaction)
Arm/Group | Part A: Dabrafenib 75 mg + Trametinib 2 mg | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg | Part C (Randomized): Dabrafenib 150 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Started | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Dose Escalation and Expansion)
Arm/Group | Part A: Dabrafenib 75 mg + Trametinib 2 mg | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg | Part C (Randomized): Dabrafenib 150 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Started | 0 | 6 | 23 | 27 | 94 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 6 | 23 | 27 | 94 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 4 | 18 | 21 | 68 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study closed/terminated | 0 | 0 | 3 | 2 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C (Phase II: Randomized Phase)
Arm/Group | Part A: Dabrafenib 75 mg + Trametinib 2 mg | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg | Part C (Randomized): Dabrafenib 150 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Started | 0 | 0 | 0 | 0 | 0 | 54 | 54 | 54 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 54 | 54 | 54 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 44 | 34 | 39 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Study closed/terminated | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 11 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C (Phase II: Crossover Phase [CP])
Arm/Group | Part A: Dabrafenib 75 mg + Trametinib 2 mg | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg | Part C (Randomized): Dabrafenib 150 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study closed/terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Period: Part D (HPMC Capsules)
Arm/Group | Part A: Dabrafenib 75 mg + Trametinib 2 mg | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg | Part C (Randomized): Dabrafenib 150 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 16 | 43 | 39
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 16 | 43 | 39
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 12 | 28 | 26
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Study closed/terminated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 10 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part C: Dabrafenib 150 mg: Participants received dabrafenib 150 mg gelatin capsules BID.
- Part C: Dabrafenib 150 mg + Trametinib 1 mg: Participants received dabrafenib 150 mg gelatin capsules BID and trametinib 1 mg tablets QD.
- Part C: Dabrafenib 150 mg + Trametinib 2 mg: Participants received dabrafenib 150 mg gelatin capsules BID and trametinib 2 mg tablets QD.
- Total: Total of all reporting groups
Arm/Group | Part A: Dabrafenib 75 mg + Trametinib 2 mg | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg | Total
Number analyzed (Participants) | 8 | 6 | 23 | 27 | 94 | 54 | 54 | 54 | 12 | 16 | 43 | 39 | 430
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (16.04) | 48.2 (7.28) | 54.2 (13.24) | 52.2 (12.09) | 52.4 (12.99) | 51.8 (15.19) | 49.9 (14.70) | 55.9 (11.85) | 51.8 (12.39) | 53.1 (17.04) | 52.8 (14.57) | 56.7 (14.08) | 52.8 (13.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 10 | 12 | 56 | 25 | 24 | 20 | 6 | 8 | 18 | 14 | 197
  Male | 6 | 4 | 13 | 15 | 38 | 29 | 30 | 34 | 6 | 8 | 25 | 25 | 233
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 7 | 6 | 22 | 26 | 92 | 52 | 54 | 53 | 12 | 16 | 43 | 39 | 407
  Asian | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Missing | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part A: Maximum Plasma Concentration (Cmax) of a Single Dose of Dabrafenib Administered Alone and in Combination With Trametnib
Description: Blood samples for PK analysis of dabrafenib and its the metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) were obtained at pre-dose and at 1, 2, 3, 4, 6, 8, 10, and 24 hours after dabrafenib administration. From the plasma concentration-time curve, the PK parameter Cmax was determined by standard non-compartmental analysis using WinNonlin. Cmax data are reported as geometric least squares means.
Time Frame: Day 15
Population: Pharmacokinetic (PK) Population: all participants who received at least one dose of either dabrafenib or trametinib and for whom a PK sample was obtained and analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter (ng/mL)
Groups:
- Part A: Dabrafenib 75 mg: Participants received a single dose of dabrafenib 75 mg gelatin capsules alone on Day 1.
Arm/Group | Part A: Dabrafenib 75 mg | Part A: Dabrafenib 75 mg + Trametinib 2 mg
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter (ng/mL)
  GSK2118436 | 509 [379 to 685] | 524 [390 to 705]
  GSK2285403 | 259 [190 to 352] | 255 [196 to 331]
  GSK2298683 | 724 [595 to 879] | 747 [587 to 951]
  GSK2167542 | 8.37 [4.82 to 14.5] | 8.16 [5.68 to 11.7]
Statistical Analysis 1: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — Cmax of dabrafenib was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = 1.03, 90% CI 2-sided [0.79 to 1.34] — Geometric mean ratio (Day 15 Cmax/Day 1 Cmax) and 90% confidence interval for dabrafenib were calculated
Statistical Analysis 2: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — Cmax of GSK2285403 was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = .99, 90% CI 2-sided [0.78 to 1.25] — Geometric mean ratio (Day 15 Cmax/Day 1 Cmax) and 90% confidence interval for GSK2285403 were calculated
Statistical Analysis 3: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — Cmax of GSK2298683 was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = 1.03, 90% CI 2-sided [0.84 to 1.27] — Geometric mean ratio (Day 15 Cmax/Day 1 Cmax) and 90% confidence interval for GSK2298683 were calculated
Statistical Analysis 4: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — Cmax of GSK2167542 was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = .98, 90% CI 2-sided [0.66 to 1.45] — Geometric mean ratio (Day 15 Cmax/Day 1 Cmax) and 90% confidence interval for GSK2167542 were calculated

2. Primary Outcome: Part A: AUC (0-t) and AUC (0-inf) of Dabrafenib and Its Metabolites
Description: Blood samples for PK analysis of dabrafenib and its metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) were obtained at pre-dose and at 1, 2, 3, 4, 6, 8, 10, and 24 hours after dabrafenib administration. AUC is defined as the area under the dabrafenib concentration-time curve as a measure of drug exposure. AUC (0-inf) is defined as the area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time. AUC (0-t) is defined as area under the concentration-time curve from time zero (pre-dose) to the last time of quantifiable concentration. Date are reported as geometric least square means.
Time Frame: Day 15
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hour/mL (ng*hr/mL)
Arm/Group | Part A: Dabrafenib 75 mg | Part A: Dabrafenib 75 mg + Trametinib 2 mg
Number analyzed (Participants) | 8 | 8
ng*hour/mL (ng*hr/mL)
  GSK2118436 AUC (0-t) | 2734 [2205 to 3390] | 2751 [2219 to 3411]
  GSK2118436 AUC (0-inf) | 3128 [2578 to 3797] | 2949 [2445 to 3556]
  GSK2285403 AUC (0-t) | 2232 [1684 to 2959] | 2287 [1899 to 2753]
  GSK2285403 AUC (0-inf) | 2819 [2231 to 3562] | 2497 [2097 to 2974]
  GSK2298683 AUC (0-t) | 12761 [10347 to 15738] | 13053 [10475 to 16266]
  GSK2298683 AUC (0-inf): number analyzed (Participants) | 0 | 0
  GSK2167542 AUC (0-t) | 270 [188 to 390] | 276 [230 to 332]
  GSK2167542 AUC (0-inf): number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — AUC(0-t) of dabrafenib was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = 1.01, 90% CI 2-sided [0.85 to 1.19] — Geometric mean ratio (Day 15 AUC(0-inf)/ Day 1 AUC(0-inf)) and 90% confidence interval for dabrafenib were calculated
Statistical Analysis 2: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — AUC(0-inf) of dabrafenib was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = 0.94, 90% CI 2-sided [0.82 to 1.08] — Geometric mean ratio (Day 15 AUC(0-inf)/ Day 1 AUC(0-inf)) and 90% confidence interval for dabrafenib were calculated
Statistical Analysis 3: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — AUC(0-t) of GSK2285403 was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = 1.02, 90% CI 2-sided [0.84 to 1.25] — Geometric mean ratio (Day 15 AUC(0-t)/ Day 1 AUC(0-t)) and 90% confidence interval for GSK2285403 were calculated
Statistical Analysis 4: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — AUC(0-inf) of GSK2285403 was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = 0.92, 90% CI 2-sided [0.81 to 1.03] — Geometric mean ratio (Day 15 AUC(0-inf)/ Day 1 AUC(0-inf)) and 90% confidence interval for GSK2285403 were calculated
Statistical Analysis 5: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — AUC(0-t) of GSK2298683 was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = 1.02, 90% CI 2-sided [0.81 to 1.29] — Geometric mean ratio (Day 15 AUC(0-t)/ Day 1 AUC(0-t)) and 90% confidence interval for GSK2298683 were calculated
Statistical Analysis 6: Comparison: Part A: Dabrafenib 75 mg vs Part A: Dabrafenib 75 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — AUC(0-t) of GSK2167542 was log e transformed and analyzed by a linear mixed effect model with fixed effect for treatment (dabrafenib alone and combined with trametinib) and participant as a random effect. Geometric mean ratio (Day 15/Day 1) and 90% confidence interval were provided; Geometric Mean Ratio = 1.02, 90% CI 2-sided [0.76 to 1.37] — Geometric mean ratio (Day 15 AUC(0-t)/ Day 1 AUC(0-t)) and 90% confidence interval for GSK2167542 were calculated

3. Primary Outcome: Part B: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 8 years)
Population: All Treated Participants (ATP) Population: all participants who received at least one dose of either dabrafenib or trametinib
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 23 | 27 | 94
Participants
  Any AE | 6 | 23 | 27 | 93
  Any SAE | 1 | 15 | 14 | 55

4. Primary Outcome: Part B: Number of Participants With Worst-case Chemistry Toxicity Grade Change From Baseline
Description: Clinical Chemistry parameters were summarized according to National Cancer Institutes (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade, version 4.0. Grade 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to Grade 3 or Grade 4 occurred. Participants with missing Baseline Grade were assumed to have Baseline Grade of 0. All increases were an increase in grade from Baseline. Only descriptive analysis.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 8 years)
Population: All Treated Participants (ATP) Population. Only participants with lab values at the specified planned time were considered.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 23 | 27 | 94
Participants
  Albumin: number analyzed (Participants) | 0 | 0 | 1 | 3
  Albumin: Increase to Grade 3 | 0 | 0 | 1 | 3
  Albumin: Increase to Grade 4 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: number analyzed (Participants) | 1 | 2 | 1 | 10
  Alkaline Phosphatase: Increase to Grade 3 | 1 | 2 | 1 | 10
  Alkaline Phosphatase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Alanine Amino Transferase: number analyzed (Participants) | 0 | 0 | 1 | 2
  Alanine Amino Transferase: Increase to Grade 3 | 0 | 0 | 1 | 2
  Alanine Amino Transferase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Amylase: number analyzed (Participants) | 0 | 0 | 0 | 0
  Amylase: Increase to Grade 3 | 0 | 0 | 0 | 0
  Amylase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Aspartate Amino Transferase: number analyzed (Participants) | 0 | 0 | 1 | 5
  Aspartate Amino Transferase: Increase to Grade 3 | 0 | 0 | 1 | 5
  Aspartate Amino Transferase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Total Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 2
  Total Bilirubin: Increase to Grade 3 | 0 | 0 | 0 | 2
  Total Bilirubin: Increase to Grade 4 | 0 | 0 | 0 | 0
  Calcium (Hypercalcemia): number analyzed (Participants) | 0 | 0 | 0 | 0
  Calcium (Hypercalcemia): Increase to Grade 3 | 0 | 0 | 0 | 0
  Calcium (Hypercalcemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Calcium (Hypocalcemia): number analyzed (Participants) | 0 | 0 | 1 | 2
  Calcium (Hypocalcemia): Increase to Grade 3 | 0 | 0 | 1 | 1
  Calcium (Hypocalcemia): Increase to Grade 4 | 0 | 0 | 0 | 1
  Creatine Kinase: number analyzed (Participants) | 0 | 0 | 0 | 0
  Creatine Kinase: Increase to Grade 3 | 0 | 0 | 0 | 0
  Creatine Kinase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Creatinine: number analyzed (Participants) | 0 | 0 | 1 | 0
  Creatinine: Increase to Grade 3 | 0 | 0 | 0 | 0
  Creatinine: Increase to Grade 4 | 0 | 0 | 1 | 0
  Gamma Glutamyl Transferase: number analyzed (Participants) | 1 | 0 | 3 | 13
  Gamma Glutamyl Transferase: Increase to Grade 3 | 1 | 0 | 3 | 13
  Gamma Glutamyl Transferase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Glucose (Hyperglycemia): number analyzed (Participants) | 0 | 2 | 2 | 5
  Glucose (Hyperglycemia): Increase to Grade 3 | 0 | 2 | 2 | 5
  Glucose (Hyperglycemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Glucose (Hypoglycemia): number analyzed (Participants) | 0 | 0 | 0 | 1
  Glucose (Hypoglycemia): Increase to Grade 3 | 0 | 0 | 0 | 1
  Glucose (Hypoglycemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Potassium (Hyperkalemia): number analyzed (Participants) | 0 | 0 | 0 | 1
  Potassium (Hyperkalemia): Increase to Grade 3 | 0 | 0 | 0 | 1
  Potassium (Hyperkalemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Potassium (Hypokalemia): number analyzed (Participants) | 0 | 0 | 1 | 4
  Potassium (Hypokalemia): Increase to Grade 3 | 0 | 0 | 1 | 4
  Potassium (Hypokalemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Lipase: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lipase: Increase to Grade 3 | 0 | 0 | 0 | 0
  Lipase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Magnesium (Hypermagnesemia): number analyzed (Participants) | 0 | 0 | 0 | 0
  Magnesium (Hypermagnesemia): Increase to Grade 3 | 0 | 0 | 0 | 0
  Magnesium (Hypermagnesemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Magnesium (Hypomagnesemia): number analyzed (Participants) | 0 | 0 | 0 | 0
  Magnesium (Hypomagnesemia): Increase to Grade 3 | 0 | 0 | 0 | 0
  Magnesium (Hypomagnesemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Sodium (Hypernatremia): number analyzed (Participants) | 0 | 0 | 0 | 0
  Sodium (Hypernatremia): Increase to Grade 3 | 0 | 0 | 0 | 0
  Sodium (Hypernatremia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Sodium (Hyponatremia): number analyzed (Participants) | 0 | 2 | 7 | 12
  Sodium (Hyponatremia): Increase to Grade 3 | 0 | 2 | 7 | 12
  Sodium (Hyponatremia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Blood pH: number analyzed (Participants) | 0 | 0 | 0 | 0
  Blood pH: Increase to Grade 3 | 0 | 0 | 0 | 0
  Blood pH: Increase to Grade 4 | 0 | 0 | 0 | 0
  Phosphorus inorganic: number analyzed (Participants) | 0 | 2 | 6 | 4
  Phosphorus inorganic: Increase to Grade 3 | 0 | 2 | 6 | 4
  Phosphorus inorganic: Increase to Grade 4 | 0 | 0 | 0 | 0
  Uric acid: number analyzed (Participants) | 1 | 0 | 0 | 1
  Uric acid: Increase to Grade 3 | 0 | 0 | 0 | 0
  Uric acid: Increase to Grade 4 | 1 | 0 | 0 | 1

5. Primary Outcome: Part B: Number of Participants With Worst-case Chemistry Change From Baseline With Respect to Normal Range
Description: For Clinical Chemistry parameters that were not graded according to NCI CTCAE criteria, changes above (High) and below (Low) the normal range were evaluated. Participants with missing Baseline were assumed to be within normal range. Participants were counted twice if the subject "Decreased to Low" and Increase to High" during the post-baseline period. Only descriptive analysis.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 8 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 23 | 27 | 94
Participants
  Direct Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0
  Direct Bilirubin: Decrease to Low | 0 | 0 | 0 | 0
  Direct Bilirubin: Increase to High | 0 | 0 | 0 | 0
  Indirect Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0
  Indirect Bilirubin: Decrease to Low | 0 | 0 | 0 | 0
  Indirect Bilirubin: Increase to High | 0 | 0 | 0 | 0
  Creatine Kinase MB mass: number analyzed (Participants) | 0 | 0 | 0 | 0
  Creatine Kinase MB mass: Decrease to Low | 0 | 0 | 0 | 0
  Creatine Kinase MB mass: Increase to High | 0 | 0 | 0 | 0
  Chloride: number analyzed (Participants) | 2 | 15 | 18 | 55
  Chloride: Decrease to Low | 0 | 4 | 10 | 39
  Chloride: Increase to High | 2 | 11 | 8 | 16
  Carbon dioxide content/Bicarbonate: number analyzed (Participants) | 4 | 11 | 17 | 41
  Carbon dioxide content/Bicarbonate: Decrease to Low | 1 | 4 | 6 | 16
  Carbon dioxide content/Bicarbonate: Increase to High | 3 | 7 | 11 | 25
  Creatinine clearance: number analyzed (Participants) | 4 | 9 | 15 | 27
  Creatinine clearance: Decrease to Low | 2 | 4 | 10 | 19
  Creatinine clearance: Increase to High | 2 | 5 | 5 | 8
  Lactate dehydrogenase: number analyzed (Participants) | 5 | 11 | 12 | 39
  Lactate dehydrogenase: Decrease to Low | 1 | 2 | 1 | 4
  Lactate dehydrogenase: Increase to High | 4 | 9 | 11 | 35
  Total protein: number analyzed (Participants) | 3 | 12 | 11 | 37
  Total protein: Decrease to Low | 0 | 10 | 10 | 30
  Total protein: Increase to High | 3 | 2 | 1 | 7
  Troponin I: number analyzed (Participants) | 0 | 0 | 0 | 0
  Troponin I: Decrease to Low | 0 | 0 | 0 | 0
  Troponin I: Increase to High | 0 | 0 | 0 | 0
  Trponin T: number analyzed (Participants) | 0 | 0 | 0 | 0
  Trponin T: Decrease to Low | 0 | 0 | 0 | 0
  Trponin T: Increase to High | 0 | 0 | 0 | 0
  Urea/BUN: number analyzed (Participants) | 3 | 14 | 19 | 47
  Urea/BUN: Decrease to Low | 2 | 4 | 3 | 17
  Urea/BUN: Increase to High | 1 | 10 | 16 | 30

6. Primary Outcome: Part B: Number of Participants With Worst-case Hematology Toxicity Grade Change From Baseline
Description: Hematology parameters were summarized according to National Cancer Institutes (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade, version 4.0. Grade 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to Grade 3 or Grade 4 occurred. Participants with missing Baseline Grade were assumed to have Baseline Grade of 0. All increases were an increase in grade from Baseline. Only descriptive analysis.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 8 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 23 | 27 | 94
Participants
  Hemoglobin (Increased): number analyzed (Participants) | 0 | 0 | 0 | 0
  Hemoglobin (Increased): Increase to Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin (Increased): Increase to Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin (Anemia): number analyzed (Participants) | 0 | 0 | 3 | 10
  Hemoglobin (Anemia): Increase to Grade 3 | 0 | 0 | 3 | 10
  Hemoglobin (Anemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Lymphocytes (Increased): number analyzed (Participants) | 0 | 0 | 0 | 0
  Lymphocytes (Increased): Increase to Grade 3 | 0 | 0 | 0 | 0
  Lymphocytes (Increased): Increase to Grade 4 | 0 | 0 | 0 | 0
  Lymphocytes (Decreased): number analyzed (Participants) | 0 | 8 | 8 | 24
  Lymphocytes (Decreased): Increase to Grade 3 | 0 | 7 | 4 | 19
  Lymphocytes (Decreased): Increase to Grade 4 | 0 | 1 | 4 | 5
  Total Neutrophils: number analyzed (Participants) | 1 | 3 | 3 | 10
  Total Neutrophils: Increase to Grade 3 | 1 | 3 | 3 | 10
  Total Neutrophils: Increase to Grade 4 | 0 | 0 | 0 | 0
  Platelet Count: number analyzed (Participants) | 0 | 0 | 2 | 2
  Platelet Count: Increase to Grade 3 | 0 | 0 | 2 | 1
  Platelet Count: Increase to Grade 4 | 0 | 0 | 0 | 1
  White Blood Cell Count: number analyzed (Participants) | 0 | 2 | 4 | 8
  White Blood Cell Count: Increase to Grade 3 | 0 | 2 | 4 | 8
  White Blood Cell Count: Increase to Grade 4 | 0 | 0 | 0 | 0

7. Primary Outcome: Part B: Number of Participants With Worst-case Hematology Change From Baseline With Respect to Normal Range
Description: For Hematology parameters that were not graded according to NCI CTCAE criteria, changes above (High) and below (Low) the normal range were evaluated. Participants with missing Baseline were assumed to be within normal range. Participants were counted twice if the subject "Decreased to Low" and Increase to High" during the post-baseline period. Only descriptive analysis.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 8 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 23 | 27 | 94
Participants
  Basophils: number analyzed (Participants) | 0 | 2 | 4 | 9
  Basophils: Decrease to Low | 0 | 0 | 0 | 2
  Basophils: Increase to High | 0 | 2 | 4 | 7
  Eosinophils: number analyzed (Participants) | 1 | 10 | 13 | 39
  Eosinophils: Decrease to Low | 1 | 5 | 6 | 28
  Eosinophils: Increase to High | 0 | 5 | 7 | 11
  Hematocrit: number analyzed (Participants) | 1 | 5 | 9 | 26
  Hematocrit: Decrease to Low | 1 | 5 | 7 | 24
  Hematocrit: Increase to High | 0 | 0 | 2 | 2
  Mean Corpuscle Hemoglobin concentration: number analyzed (Participants) | 2 | 10 | 16 | 34
  Mean Corpuscle Hemoglobin concentration: Decrease to Low | 0 | 6 | 11 | 21
  Mean Corpuscle Hemoglobin concentration: Increase to High | 2 | 4 | 5 | 13
  Mean Corpuscle Hemoglobin: number analyzed (Participants) | 0 | 9 | 14 | 23
  Mean Corpuscle Hemoglobin: Decrease to Low | 0 | 6 | 8 | 12
  Mean Corpuscle Hemoglobin: Increase to High | 0 | 3 | 6 | 11
  Mean Corpuscle Volume: number analyzed (Participants) | 2 | 7 | 10 | 18
  Mean Corpuscle Volume: Decrease to Low | 1 | 5 | 6 | 13
  Mean Corpuscle Volume: Increase to High | 1 | 2 | 4 | 5
  Monocytes: number analyzed (Participants) | 3 | 12 | 19 | 51
  Monocytes: Decrease to Low | 2 | 8 | 10 | 21
  Monocytes: Increase to High | 1 | 4 | 9 | 30
  Red Blood Cell count: number analyzed (Participants) | 1 | 9 | 6 | 27
  Red Blood Cell count: Decrease to Low | 1 | 9 | 5 | 25
  Red Blood Cell count: Increase to High | 0 | 0 | 1 | 2
  Reticulocytes: number analyzed (Participants) | 4 | 8 | 11 | 9
  Reticulocytes: Decrease to Low | 2 | 1 | 5 | 3
  Reticulocytes: Increase to High | 2 | 7 | 6 | 6

8. Primary Outcome: Part B: Number of Participants With the Indicated Worst-case Change From Baseline in Heart Rate and Blood Pressure
Description: Blood pressure and heart rate were summarized according to NCI CTCAE grade, version 4.0. Grade 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to G3 or G4 occurred. Blood pressure measurement included systolic blood pressure (SBP, millimeters of mercury [mmHg]) and diastolic BP (DBP). Heart rate is the measure of heart beats per minute (bpm). Changes in heart rate, either decrease to <60 bpm, change to normal or no change, or increase to >100 bpm are presented.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 8 years)
Population: ATP Population
Measure: Number; unit: Participants
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 23 | 27 | 78
Participants
  Heart rate, Decrease to <60 bpm | 1 | 2 | 5 | 15
  Heart rate, Change to normal or no change | 3 | 14 | 15 | 37
  Heart rate, Increase to >100 bpm | 2 | 7 | 8 | 26
  SBP, Increase to G3 or G4 | 0 | 2 | 3 | 8
  DBP, Increase to G3 or G4 | 0 | 1 | 3 | 4

9. Primary Outcome: Part C (Randomized): Number of Participants With BRAF Mutant Metastatic Melanoma With Best Overall Response as Assessed by the Investigator
Description: Best overall response is defined as complete response (CR: the disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeters [mm] in the short axis.) or partial reponse (PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). Participants with unknown or missing responses were considered as non-responders. To be assigned a status of PR or CR, a confirmatory disease assessment should have been performed no less than 28 days after the criteria for response were first met. Response was evaluated by an investigator as per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
Time Frame: From the first dose of study medication to the first documented evidence of a confirmed complete response or partial response (up to approximately 7 years)
Population: Intent-to-Treat (ITT) Population: all randomized participants regardless of whether or not treatment was administered
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 54 | 54 | 54
Participants
  CR | 2 | 6 | 10
  PR | 27 | 21 | 31
Statistical Analysis 1: Comparison: Part C: Dabrafenib 150 mg vs Part C: Dabrafenib 150 mg + Trametinib 1 mg; Difference in response rate Arm2 - Arm1; Test type: Superiority or Other; Unconditional exact method = -4, 95% CI 2-sided [-23.1 to 15.9]
Statistical Analysis 2: Comparison: Part C: Dabrafenib 150 mg vs Part C: Dabrafenib 150 mg + Trametinib 2 mg; Difference in response rate Arm3 - Arm1; Test type: Superiority or Other; Unconditional exact method = 22, 95% CI 2-sided [2.5 to 40.7]

10. Primary Outcome: Part C (Randomized): Number of Participants With BRAF Mutant Metastatic Melanoma With Best Overall Response Assessed by Blinded Independent Central Review (BICR)
Description: Best overall response is defined as complete response (CR: the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or partial reponse (PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). Participants with unknown or missing responses were considered as non-responders. To be assigned a status of PR or CR, a confirmatory disease assessment should have been performed no less than 28 days after the criteria for response were first met. Response was evaluated by BICR as per RECIST, version 1.1.
Time Frame: From the first dose of study medication to the first documented evidence of a confirmed complete response or partial response (up to approximately 19 months)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 54 | 54 | 54
Participants
  CR | 4 | 4 | 7
  PR | 21 | 18 | 26
Statistical Analysis 1: Comparison: Part C: Dabrafenib 150 mg vs Part C: Dabrafenib 150 mg + Trametinib 1 mg; Difference in response rate Arm2- Arm1; Test type: Superiority or Other; Unconditional exact method = -6, 95% CI 2-sided [-24.9 to 14.1]
Statistical Analysis 2: Comparison: Part C: Dabrafenib 150 mg vs Part C: Dabrafenib 150 mg + Trametinib 2 mg; Difference in response rate Arm3 - Arm1; Test type: Superiority or Other; Unconditional exact method = 15, 95% CI 2-sided [-4.9 to 33.7]

11. Primary Outcome: Part C (Crossover): Number of Participants With BRAF Mutant Metastatic Melanoma With Best Overall Response as Assessed by the Investigator
Description: Best overall response is defined as complete response (CR: the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or partial reponse (PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). Participants with unknown or missing responses were considered as non-responders. To be assigned a status of PR or CR, a confirmatory disease assessment should have been performed no less than 28 days after the criteria for response were first met. Response was evaluated by an investigator as per RECIST, version 1.1.
Time Frame: as for outcome 9
Population: Crossover Population: participants who were randomized to and received at least one dose of dabrafenib monotherapy, and who elected to crossover to combination therapy following disease progression while on monotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 45
Participants
  CR | 1
  PR | 5
Statistical Analysis 1: Comparison: Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg; Test type: Superiority or Other; Response rate = 6, 95% CI 2-sided [5.1 to 26.8]

12. Primary Outcome: Part C (Randomized): Progression-free Survival (PFS) as Assessed by the Investigator
Description: PFS is defined as the interval between the date of randomization and the earliest date of PD or death due to any cause. PD was based on radiographic or photographic evidence, and assessments were made by the investigator according to RECIST, version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. Participants who received anti-cancer therapy prior to the date of documented events, were censored at the last adequate assessment prior to the initiation of therapy. If the participant did not had a documented date of events, PFS and survival were censored at the date of the last adequate assessment.
Time Frame: From the date of randomization to the earliest date of disease progression (PD) or death due to any cause (up to approximately 7 years)
Population: ITT Population
Measure: Median (Full Range); unit: Months
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 54 | 54 | 54
Months | 5.8 [4.3 to 7.4] | 9.2 [5.7 to 11.0] | 9.4 [7.6 to 16.6]
Statistical Analysis 1: Comparison: Part C: Dabrafenib 150 mg vs Part C: Dabrafenib 150 mg + Trametinib 1 mg; Test type: Superiority or Other; p = 0.0048, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.38 to 0.87] — HRs were estimated using the Pike estimator
Statistical Analysis 2: Comparison: Part C: Dabrafenib 150 mg vs Part C: Dabrafenib 150 mg + Trametinib 2 mg; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.29 to 0.68] — HRs were estimated using the Pike estimator

13. Primary Outcome: Part C (Crossover): Progression-free Survival (PFS) as Assessed by the Investigator
Description: PFS is defined as the interval between the first dose of study medication and the earliest date of PD or death due to any cause. PD was based on radiographic or photographic evidence, and assessments were made by the investigator according to RECIST, version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. Participants received anti-cancer therapy prior to the date of documented events, and censored at the last adequate assessment, prior to the initiation of therapy. If the participant did not have a documented date of events, PFS and survival were censored at the date of the last adequate assessment.
Time Frame: From the first dose of study medication to the earliest date of disease progression (PD) or death due to any cause (up to approximately 7 years)
Population: Crossover Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 45
Months | 3.6 [1.8 to 3.9]

14. Primary Outcome: Part C (Randomized): Progression-free Survival (PFS) as Assessed by the Blinded Independent Central Review (BICR)
Description: PFS is defined as the interval between the date of randomization and the earliest date of PD or death due to any cause. PD was based on radiographic or photographic evidence, and assessments were made by the BICR according to RECIST, version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. Participants who received anti-cancer therapy prior to the date of documented events, were censored at the last adequate assessment prior to the initiation of therapy. If the participant did not had a documented date of events, PFS and survival were censored at the date of the last adequate assessment
Time Frame: From the date of randomization to the earliest date of disease progression (PD) or death due to any cause (up to approximately 19 months)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 54 | 54 | 54
Months | 7.3 [5.5 to 9.4] | 8.3 [5.6 to 11.3] | 9.2 [7.6 to NA] — NA: Not estimable due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Part C: Dabrafenib 150 mg vs Part C: Dabrafenib 150 mg + Trametinib 1 mg; Test type: Superiority or Other; p = 0.1667, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.45 to 1.18] — HRs were estimated using the Pike estimator
Statistical Analysis 2: Comparison: Part C: Dabrafenib 150 mg vs Part C: Dabrafenib 150 mg + Trametinib 2 mg; Test type: Superiority or Other; p = 0.0119, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.32 to 0.90] — HRs were estimated using the Pike estimator

15. Primary Outcome: Part C (Randomized): Duration of Response as Assessed by the Investigator and Blinded Independent Central Review (BICR)
Description: Duration of response for participants with either a CR (the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]) is defined as the time from the first documented evidence of a PR or CR until the first documented sign of disease progression (PD) or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: First documented evidence of PR or CR until the date of the first documented sign of disease progression or the date of death due to any cause (up to approximately 19 months)
Population: ITT Population. Only those participants who had a CR or PR were analyzed for duration of response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 54 | 54 | 54
Months
  Investigator assessed: number analyzed (Participants) | 29 | 27 | 41
  Investigator assessed | 5.6 [3.9 to 7.4] | 11.1 [7.4 to 13.2] | 10.5 [7.4 to 19.2]
  BICR assessed: number analyzed (Participants) | 25 | 22 | 33
  BICR assessed | 7.6 [4.7 to NA] — NA: Not estimable due to insufficient number of participants with events | 9.5 [5.6 to NA] — NA: Not estimable due to insufficient number of participants with events | NA [6.7 to NA] — NA: Not estimable due to insufficient number of participants with events

16. Primary Outcome: Part C (Randomized): Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event of possible drug-induced liver injury.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: ATP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants
  Any AE | 53 | 53 | 55
  Any SAE | 15 | 24 | 39

17. Primary Outcome: Part C (Randomized): Number of Participants With Worst-case Chemistry Toxicity Grade Change From Baseline
Description: as for outcome 4
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants
  Albumin: number analyzed (Participants) | 0 | 1 | 1
  Albumin: Increase to Grade 3 | 0 | 1 | 1
  Albumin: Increase to Grade 4 | 0 | 0 | 0
  Alkaline Phosphatase: number analyzed (Participants) | 0 | 3 | 2
  Alkaline Phosphatase: Increase to Grade 3 | 0 | 3 | 2
  Alkaline Phosphatase: Increase to Grade 4 | 0 | 0 | 0
  Alanine Amino Transferase: number analyzed (Participants) | 0 | 2 | 2
  Alanine Amino Transferase: Increase to Grade 3 | 0 | 2 | 2
  Alanine Amino Transferase: Increase to Grade 4 | 0 | 0 | 0
  Aspartate Amino Transferase: number analyzed (Participants) | 0 | 1 | 3
  Aspartate Amino Transferase: Increase to Grade 3 | 0 | 1 | 3
  Aspartate Amino Transferase: Increase to Grade 4 | 0 | 0 | 0
  Total Bilirubin: number analyzed (Participants) | 0 | 2 | 0
  Total Bilirubin: Increase to Grade 3 | 0 | 2 | 0
  Total Bilirubin: Increase to Grade 4 | 0 | 0 | 0
  Calcium (Hypercalcemia): number analyzed (Participants) | 0 | 1 | 0
  Calcium (Hypercalcemia): Increase to Grade 3 | 0 | 0 | 0
  Calcium (Hypercalcemia): Increase to Grade 4 | 0 | 1 | 0
  Calcium (Hypocalcemia): number analyzed (Participants) | 0 | 0 | 0
  Calcium (Hypocalcemia): Increase to Grade 3 | 0 | 0 | 0
  Calcium (Hypocalcemia): Increase to Grade 4 | 0 | 0 | 0
  Cholesterol: number analyzed (Participants) | 0 | 0 | 0
  Cholesterol: Increase to Grade 3 | 0 | 0 | 0
  Cholesterol: Increase to Grade 4 | 0 | 0 | 0
  Creatine Kinase: number analyzed (Participants) | 0 | 1 | 0
  Creatine Kinase: Increase to Grade 3 | 0 | 0 | 0
  Creatine Kinase: Increase to Grade 4 | 0 | 1 | 0
  Creatinine: number analyzed (Participants) | 0 | 1 | 3
  Creatinine: Increase to Grade 3 | 0 | 1 | 2
  Creatinine: Increase to Grade 4 | 0 | 0 | 1
  Gamma Glutamyl Transferase: number analyzed (Participants) | 1 | 11 | 8
  Gamma Glutamyl Transferase: Increase to Grade 3 | 1 | 11 | 7
  Gamma Glutamyl Transferase: Increase to Grade 4 | 0 | 0 | 1
  Glucose (Hyperglycemia): number analyzed (Participants) | 1 | 4 | 6
  Glucose (Hyperglycemia): Increase to Grade 3 | 1 | 4 | 6
  Glucose (Hyperglycemia): Increase to Grade 4 | 0 | 0 | 0
  Glucose (Hypoglycemia): number analyzed (Participants) | 0 | 0 | 0
  Glucose (Hypoglycemia): Increase to Grade 3 | 0 | 0 | 0
  Glucose (Hypoglycemia): Increase to Grade 4 | 0 | 0 | 0
  Potassium (Hyperkalemia): number analyzed (Participants) | 2 | 0 | 1
  Potassium (Hyperkalemia): Increase to Grade 3 | 2 | 0 | 1
  Potassium (Hyperkalemia): Increase to Grade 4 | 0 | 0 | 0
  Potassium (Hypokalemia): number analyzed (Participants) | 3 | 1 | 2
  Potassium (Hypokalemia): Increase to Grade 3 | 3 | 1 | 1
  Potassium (Hypokalemia): Increase to Grade 4 | 0 | 0 | 1
  Magnesium (Hypermagnesemia): number analyzed (Participants) | 0 | 2 | 1
  Magnesium (Hypermagnesemia): Increase to Grade 3 | 0 | 2 | 1
  Magnesium (Hypermagnesemia): Increase to Grade 4 | 0 | 0 | 0
  Magnesium (Hypomagnesemia): number analyzed (Participants) | 0 | 0 | 1
  Magnesium (Hypomagnesemia): Increase to Grade 3 | 0 | 0 | 1
  Magnesium (Hypomagnesemia): Increase to Grade 4 | 0 | 0 | 0
  Sodium (Hypernatremia): number analyzed (Participants) | 0 | 0 | 0
  Sodium (Hypernatremia): Increase to Grade 3 | 0 | 0 | 0
  Sodium (Hypernatremia): Increase to Grade 4 | 0 | 0 | 0
  Sodium (Hyponatremia): number analyzed (Participants) | 0 | 10 | 6
  Sodium (Hyponatremia): Increase to Grade 3 | 0 | 10 | 6
  Sodium (Hyponatremia): Increase to Grade 4 | 0 | 0 | 0
  Phosphorus inorganic: number analyzed (Participants) | 0 | 6 | 4
  Phosphorus inorganic: Increase to Grade 3 | 0 | 6 | 4
  Phosphorus inorganic: Increase to Grade 4 | 0 | 0 | 0
  Triglycerides: number analyzed (Participants) | 0 | 0 | 0
  Triglycerides: Increase to Grade 3 | 0 | 0 | 0
  Triglycerides: Increase to Grade 4 | 0 | 0 | 0

18. Primary Outcome: Part C (Randomized): Number of Participants With Worst-case Chemistry Change From Baseline With Respect to Normal Range
Description: as for outcome 5
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: ATP Population. Only those participants who were available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants
  Direct Bilirubin: number analyzed (Participants) | 0 | 0 | 0
  Direct Bilirubin: Decrease to Low | 0 | 0 | 0
  Direct Bilirubin: Increase to High | 0 | 0 | 0
  Creatine Kinase MB mass: number analyzed (Participants) | 0 | 1 | 0
  Creatine Kinase MB mass: Decrease to Low | 0 | 0 | 0
  Creatine Kinase MB mass: Increase to High | 0 | 1 | 0
  Chloride: number analyzed (Participants) | 18 | 38 | 36
  Chloride: Decrease to Low | 7 | 24 | 24
  Chloride: Increase to High | 11 | 14 | 12
  Carbon dioxide content/Bicarbonate: number analyzed (Participants) | 13 | 22 | 28
  Carbon dioxide content/Bicarbonate: Decrease to Low | 5 | 8 | 12
  Carbon dioxide content/Bicarbonate: Increase to High | 8 | 14 | 16
  C-Reactive protein: number analyzed (Participants) | 0 | 0 | 3
  C-Reactive protein: Decrease to Low | 0 | 0 | 0
  C-Reactive protein: Increase to High | 0 | 0 | 3
  Creatinine Clearance: number analyzed (Participants) | 14 | 27 | 20
  Creatinine Clearance: Decrease to Low | 7 | 16 | 10
  Creatinine Clearance: Increase to High | 7 | 11 | 10
  High Density Lipids, Cholesterol: number analyzed (Participants) | 0 | 0 | 0
  High Density Lipids, Cholesterol: Decrease to Low | 0 | 0 | 0
  High Density Lipids, Cholesterol: Increase to High | 0 | 0 | 0
  Lactate Dehydrogenase: number analyzed (Participants) | 5 | 27 | 34
  Lactate Dehydrogenase: Decrease to Low | 2 | 3 | 2
  Lactate Dehydrogenase: Increase to High | 3 | 24 | 32
  Low Density Lipids, Cholesterol: number analyzed (Participants) | 0 | 0 | 0
  Low Density Lipids, Cholesterol: Decrease to Low | 0 | 0 | 0
  Low Density Lipids, Cholesterol: Increase to High | 0 | 0 | 0
  Total Protein: number analyzed (Participants) | 5 | 18 | 22
  Total Protein: Decrease to Low | 4 | 10 | 19
  Total Protein: Increase to High | 1 | 8 | 3
  Troponin I: number analyzed (Participants) | 0 | 0 | 0
  Troponin I: Decrease to Low | 0 | 0 | 0
  Troponin I: Increase to High | 0 | 0 | 0
  Urea/BUN: number analyzed (Participants) | 13 | 27 | 29
  Urea/BUN: Decrease to Low | 5 | 4 | 9
  Urea/BUN: Increase to High | 8 | 23 | 20

19. Primary Outcome: Part C (Randomized): Number of Participants With Worst-case Hematology Toxicity Grade Change From Baseline
Description: Hematology parameters were summarized according to National Cancer Institutes (NCI) CTCAE grade, version 4.0. Grade 1, Mild; Grade 2, Moderate; Grade 3, Severe; Grade 4, Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase Grade 3 or Grade 4 occurred. Participants with missing Baseline Grade were assumed to have Baseline Grade of 0. All increases were an increase in grade from Baseline. Only descriptive analysis.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants
  Hemoglobin (Increased): number analyzed (Participants) | 0 | 0 | 0
  Hemoglobin (Increased): Increase to Grade 3 | 0 | 0 | 0
  Hemoglobin (Increased): Increase to Grade 4 | 0 | 0 | 0
  Hemoglobin (Anemia): number analyzed (Participants) | 0 | 4 | 2
  Hemoglobin (Anemia): Increase to Grade 3 | 0 | 4 | 2
  Hemoglobin (Anemia): Increase to Grade 4 | 0 | 0 | 0
  Lymphocytes (Increased): number analyzed (Participants) | 0 | 0 | 0
  Lymphocytes (Increased): Increase to Grade 3 | 0 | 0 | 0
  Lymphocytes (Increased): Increase to Grade 4 | 0 | 0 | 0
  Lymphocytes (Decreased): number analyzed (Participants) | 3 | 11 | 15
  Lymphocytes (Decreased): Increase to Grade 3 | 3 | 10 | 12
  Lymphocytes (Decreased): Increase to Grade 4 | 0 | 1 | 3
  Total Neutrophils: number analyzed (Participants) | 1 | 2 | 8
  Total Neutrophils: Increase to Grade 3 | 1 | 2 | 4
  Total Neutrophils: Increase to Grade 4 | 0 | 0 | 4
  Platelet Count: number analyzed (Participants) | 0 | 2 | 4
  Platelet Count: Increase to Grade 3 | 0 | 2 | 3
  Platelet Count: Increase to Grade 4 | 0 | 0 | 1
  White Blood Cell count: number analyzed (Participants) | 0 | 3 | 5
  White Blood Cell count: Increase to Grade 3 | 0 | 3 | 5
  White Blood Cell count: Increase to Grade 4 | 0 | 0 | 0

20. Primary Outcome: Part C (Randomized): Number of Participants With Worst-case Hematology Change From Baseline With Respect to Normal Range
Description: as for outcome 7
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants
  Basophils: number analyzed (Participants) | 4 | 7 | 13
  Basophils: Decrease to Low | 1 | 1 | 3
  Basophils: Increase to High | 3 | 6 | 10
  Eosinophils: number analyzed (Participants) | 5 | 22 | 17
  Eosinophils: Decrease to Low | 3 | 11 | 8
  Eosinophils: Increase to High | 2 | 11 | 9
  Hematocrit: number analyzed (Participants) | 17 | 24 | 29
  Hematocrit: Decrease to Low | 15 | 23 | 27
  Hematocrit: Increase to High | 2 | 1 | 2
  Mean Corpuscle Hemoglobin concentration: number analyzed (Participants) | 13 | 24 | 21
  Mean Corpuscle Hemoglobin concentration: Decrease to Low | 11 | 16 | 12
  Mean Corpuscle Hemoglobin concentration: Increase to High | 2 | 8 | 9
  Mean Corpuscle Hemoglobin: number analyzed (Participants) | 10 | 17 | 16
  Mean Corpuscle Hemoglobin: Decrease to Low | 6 | 11 | 8
  Mean Corpuscle Hemoglobin: Increase to High | 4 | 6 | 8
  Mean Corpuscle Volume: number analyzed (Participants) | 9 | 10 | 11
  Mean Corpuscle Volume: Decrease to Low | 8 | 5 | 7
  Mean Corpuscle Volume: Increase to High | 1 | 5 | 4
  Monocytes: number analyzed (Participants) | 22 | 34 | 26
  Monocytes: Decrease to Low | 5 | 14 | 12
  Monocytes: Increase to High | 17 | 20 | 14
  Red Blood Cell count: number analyzed (Participants) | 12 | 26 | 29
  Red Blood Cell count: Decrease to Low | 11 | 22 | 25
  Red Blood Cell count: Increase to High | 1 | 4 | 4
  Reticulocytes: number analyzed (Participants) | 0 | 1 | 7
  Reticulocytes: Decrease to Low | 0 | 1 | 2
  Reticulocytes: Increase to High | 0 | 0 | 5

21. Primary Outcome: Part C (Randomized): Number of Participants With the Indicated Worst-case Change From Baseline in Heart Rate and Blood Pressure
Description: Blood pressure were summarized according to National Cancer Institutes (NCI) CTCAE grade, version 4.0. Grade 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to G3 or G4 occurred.lood pressure measurement included systolic blood pressure (BP, milimeter of mercury [mmHg]) and diastolic BP (DBP). Worst case change from Baseline was calculated as the post-Baseline value minus the Baseline value. Heart Rate is the measure of heart beats per minute (bpm). Changes in heart rate, either decrease to <60 bpm, change to normal or no change, or increase to >100 bpm are presented.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: ATP Population
Measure: Number; unit: Participants
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 53 | 54 | 55
Participants
  Systolic BP (mmHg) , G3 or G4 | 5 | 4 | 12
  Diastolic BP (mmHg), G3 or G4 | 4 | 4 | 4
  Heart rate, Decrease to <60 bpm | 9 | 8 | 11
  Heart rate, Change to normal or no change | 34 | 30 | 28
  Heart rate, Increase to >100 bpm | 10 | 16 | 18

22. Primary Outcome: Part D (Analyte=GSK2118436): Maximum Plasma Concentration (Cmax) of a Single and Repeat Dose of Dabrafenib Alone and in Combination With Trametinib
Description: The PK parameter Cmax was assessed. Blood samples for PK analysis of dabrafenib were obtained at pre-dose Day 1 and Day 21 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours (24 hour on Day 1 only) post-dose administration. From the plasma concentration-time curve, the PK parameter tmax was determined by standard non-compartmental analysis using WinNonlin. Cmax data are reported as geometric least squares means.
Time Frame: Day 1 and Day 21
Population: PK Population: all participants who received at least one dose of either dabrafenib or trametinib and for whom a PK sample was obtained and analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15
ng/mL
  Day 1 | 1117 [914 to 1365] | 1669 [1059 to 2631] | 1227 [924 to 1764] | 2289 [1622 to 3231]
  Day 21 | 1050 [811 to 1358] | 1746 [1344 to 2269] | 1217 [895 to 1654] | 2052 [1472 to 2860]
Statistical Analysis 1: Comparison: Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg vs Part D: Dabrafenib 150 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — Following loge tranformation, Cmax of dabrafenib after repeat doses from the pooled data in Part B and D were analyzed by a linear model with the following fixed effects as categorical variables: Capsule type (Gelatin or HPMC), BRAF dose (75 or 150 mg BID), Capsule type by BRAF dose interaction, Day (Day 15 or 21), MEK dose (0, 1, 1.5 or 2 mg QD). Geometric mean ratio (HPMC/Gelatin) and the corresponding 90% CI were provided for BRAF dose level 150 mg BID; Geometric Mean Ratio = 1.51, 90% CI 2-sided [1.10 to 2.08] — Geometric mean ratio (HPMC/Gelatin) and the corresponding 90% CI were provided for BRAF dose level 150 mg BID

23. Primary Outcome: Part D (Analyte=GSK2118436): Tmax of a Single and Repeat Dose of Dabrafenib Alone and in Combination With Trametinib
Description: tmax is defined as the time of occurenceof Cmax. Blood samples for PK analysis of dabrafenib were obtained at Day 1 and Day 21 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours (24 hour on Day 1 only) post-dose administration. From the plasma concentration-time curve, the PK parameter tmax was determined by standard non-compartmental analysis using WinNonlin.
Time Frame: Day 1 and Day 21
Population: PK Population. Only participants available at the indicated timepoints were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15
Hours
  Day 1 | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 6.00] | 2.00 [1.00 to 3.00] | 1.50 [1.00 to 10.00]
  Day 21 | 1.50 [1.00 to 2.00] | 1.55 [0.98 to 3.00] | 1.75 [1.00 to 3.00] | 1.50 [1.00 to 3.00]

24. Primary Outcome: Part D (Analyte=GSK2118436): AUC (0-tau) and AUC (0-inf) of Single and Repeat Doses of Dabrafenib Alone and in Combination With Trametinib
Description: The PK parameters were determined for area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration AUC (0-tau) and from time zero (pre-dose) extrapolated to infinite time AUC (0-inf). Blood samples for PK analysis of the metabolites of dabrafenib were obtained at Day 1 and Day 21 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours (24 hour only on Day 1) post-dose administration.
Time Frame: Day 1 and Day 21
Population: PK Population. Only participants available at the indicated timepoints were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15
ng*hr/mL
  AUC (0-tau), Day 1 | 3593 [3008 to 4293] | 6507 [4288 to 9872] | 4618 [3525 to 6051] | 7331 [5355 to 10037]
  AUC (0-tau), Day 21 | 3020 [2390 to 3816] | 4663 [3511 to 6194] | 3434 [2679 to 4403] | 5886 [4608 to 7517]
  AUC (0-inf), Day 1 | 3982 [3325 to 4770] | 7291 [4830 to 11005] | 5321 [4192 to 6755] | 8152 [5860 to 11341]
  AUC (0-inf), Day 21: number analyzed (Participants) | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg vs Part D: Dabrafenib 150 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — Following loge transformation, AUC(0-tau) of dabrafenib was analyzed by a linear mixed effect model with dosing chort and day as fixed effects and subject as random effect. Based on the model, geometric mean ratio (Day 21 Dabrafenib 150 mg BID+Trametinib 2 mg QD/Day 21 Dabrafenib 150 mg BID alone) and the corresponding 90% confidence interval were provided; Geometric Mean Ratio = 1.23, 90% CI 2-sided [0.89 to 1.69] — Geometric mean ratio (Day 21 Dabrafenib 150 mg BID+Trametinib 2 mg QD/Day 21 Dabrafenib 150 mg BID alone) and the corresponding 90% confidence interval were provided
Statistical Analysis 2: Comparison: Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg vs Part D: Dabrafenib 150 mg + Trametinib 2 mg; Test type: Non-Inferiority or Equivalence — Following loge tranformation, AUC(0-tau) of dabrafenib after repeat doses from the pooled data in Part B and D were analyzed by a linear model with the following fixed effects as categorical variables: Capsule type (Gelatin or HPMC), BRAF dose (75 or 150 mg BID), Capsule type by BRAF dose interaction, Day (Day 15 or 21), MEK dose (0, 1, 1.5, 2 or 2 mg QD). Geometric mean ratio (HPMC/Gelatin) and the corresponding 90% CI were then provided for BRAF dose level 150 mg BID; Geometric Mean Ratio = 1.10, 90% CI 2-sided [0.84 to 1.44] — Geometric mean ratio (HPMC/Gelatin) and the corresponding 90% CI were provided for BRAF dose level 150 mg BID

25. Primary Outcome: Part D: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is an event for possible drug-induced liver injury.
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: ATP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 15 | 41 | 39
Participants
  Any AE | 15 | 15 | 41 | 38
  Any SAE | 8 | 11 | 29 | 30

26. Primary Outcome: Part D: Number of Participants With Worst-case Chemistry Toxicity Grade Change From Baseline
Description: as for outcome 4
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 15 | 41 | 39
Participants
  Albumin: number analyzed (Participants) | 0 | 2 | 1 | 0
  Albumin: Increase to Grade 3 | 0 | 2 | 1 | 0
  Albumin: Increase to Grade 4 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: number analyzed (Participants) | 1 | 2 | 0 | 3
  Alkaline Phosphatase: Increase to Grade 3 | 1 | 2 | 0 | 3
  Alkaline Phosphatase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Alanine Amino Transferase: number analyzed (Participants) | 2 | 0 | 2 | 1
  Alanine Amino Transferase: Increase to Grade 3 | 2 | 0 | 2 | 1
  Alanine Amino Transferase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Amylase: number analyzed (Participants) | 0 | 0 | 0 | 0
  Amylase: Increase to Grade 3 | 0 | 0 | 0 | 0
  Amylase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Aspartate Amino Transferase: number analyzed (Participants) | 2 | 0 | 3 | 3
  Aspartate Amino Transferase: Increase to Grade 3 | 2 | 0 | 3 | 3
  Aspartate Amino Transferase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Total Bilirubin: number analyzed (Participants) | 1 | 0 | 0 | 1
  Total Bilirubin: Increase to Grade 3 | 1 | 0 | 0 | 1
  Total Bilirubin: Increase to Grade 4 | 0 | 0 | 0 | 0
  Calcium (Hypercalcemia): number analyzed (Participants) | 0 | 0 | 0 | 1
  Calcium (Hypercalcemia): Increase to Grade 3 | 0 | 0 | 0 | 1
  Calcium (Hypercalcemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Calcium (Hypocalcemia): number analyzed (Participants) | 0 | 1 | 1 | 1
  Calcium (Hypocalcemia): Increase to Grade 3 | 0 | 1 | 0 | 1
  Calcium (Hypocalcemia): Increase to Grade 4 | 0 | 0 | 1 | 0
  Cholesterol: number analyzed (Participants) | 0 | 0 | 0 | 0
  Cholesterol: Increase to Grade 3 | 0 | 0 | 0 | 0
  Cholesterol: Increase to Grade 4 | 0 | 0 | 0 | 0
  Creatine Kinase: number analyzed (Participants) | 0 | 1 | 2 | 0
  Creatine Kinase: Increase to Grade 3 | 0 | 1 | 2 | 0
  Creatine Kinase: Increase to Grade 4 | 0 | 0 | 0 | 0
  Creatinine: number analyzed (Participants) | 0 | 0 | 1 | 0
  Creatinine: Increase to Grade 3 | 0 | 0 | 1 | 0
  Creatinine: Increase to Grade 4 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase: number analyzed (Participants) | 4 | 3 | 6 | 5
  Gamma Glutamyl Transferase: Increase to Grade 3 | 3 | 1 | 6 | 5
  Gamma Glutamyl Transferase: Increase to Grade 4 | 1 | 2 | 0 | 0
  Glucose (Hyperglycemia): number analyzed (Participants) | 1 | 2 | 4 | 1
  Glucose (Hyperglycemia): Increase to Grade 3 | 1 | 2 | 4 | 1
  Glucose (Hyperglycemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Glucose (Hypoglycemia): number analyzed (Participants) | 0 | 0 | 0 | 0
  Glucose (Hypoglycemia): Increase to Grade 3 | 0 | 0 | 0 | 0
  Glucose (Hypoglycemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Potassium (Hyperkalemia): number analyzed (Participants) | 0 | 0 | 1 | 0
  Potassium (Hyperkalemia): Increase to Grade 3 | 0 | 0 | 1 | 0
  Potassium (Hyperkalemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Potassium (Hypokalemia): number analyzed (Participants) | 0 | 1 | 2 | 2
  Potassium (Hypokalemia): Increase to Grade 3 | 0 | 1 | 1 | 2
  Potassium (Hypokalemia): Increase to Grade 4 | 0 | 0 | 1 | 0
  Lipase: number analyzed (Participants) | 0 | 2 | 0 | 1
  Lipase: Increase to Grade 3 | 0 | 0 | 0 | 0
  Lipase: Increase to Grade 4 | 0 | 2 | 0 | 1
  Magnesium (Hypermagnesemia): number analyzed (Participants) | 0 | 0 | 0 | 0
  Magnesium (Hypermagnesemia): Increase to Grade 3 | 0 | 0 | 0 | 0
  Magnesium (Hypermagnesemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Magnesium (Hypomagnesemia): number analyzed (Participants) | 0 | 0 | 1 | 0
  Magnesium (Hypomagnesemia): Increase to Grade 3 | 0 | 0 | 1 | 0
  Magnesium (Hypomagnesemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Sodium (Hypernatremia): number analyzed (Participants) | 0 | 0 | 0 | 0
  Sodium (Hypernatremia): Increase to Grade 3 | 0 | 0 | 0 | 0
  Sodium (Hypernatremia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Sodium (Hyponatremia): number analyzed (Participants) | 1 | 4 | 6 | 6
  Sodium (Hyponatremia): Increase to Grade 3 | 1 | 4 | 5 | 5
  Sodium (Hyponatremia): Increase to Grade 4 | 0 | 0 | 1 | 1
  Phosphorus inorganic: number analyzed (Participants) | 0 | 0 | 3 | 2
  Phosphorus inorganic: Increase to Grade 3 | 0 | 0 | 3 | 2
  Phosphorus inorganic: Increase to Grade 4 | 0 | 0 | 0 | 0
  Triglycerides: number analyzed (Participants) | 0 | 0 | 0 | 0
  Triglycerides: Increase to Grade 3 | 0 | 0 | 0 | 0
  Triglycerides: Increase to Grade 4 | 0 | 0 | 0 | 0
  Uric acid: number analyzed (Participants) | 0 | 0 | 2 | 0
  Uric acid: Increase to Grade 3 | 0 | 0 | 0 | 0
  Uric acid: Increase to Grade 4 | 0 | 0 | 2 | 0

27. Primary Outcome: Part D: Number of Participants With Worst-case Chemistry Change From Baseline With Respect to Normal Range
Description: as for outcome 5
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 15 | 41 | 39
Participants
  Direct Bilirubin: number analyzed (Participants) | 0 | 0 | 0 | 0
  Direct Bilirubin: Decrease Low | 0 | 0 | 0 | 0
  Direct Bilirubin: Increase to High | 0 | 0 | 0 | 0
  Creatine Kinase MB mass: number analyzed (Participants) | 0 | 0 | 1 | 0
  Creatine Kinase MB mass: Decrease Low | 0 | 0 | 0 | 0
  Creatine Kinase MB mass: Increase to High | 0 | 0 | 1 | 0
  Chloride: number analyzed (Participants) | 9 | 11 | 25 | 34
  Chloride: Decrease Low | 7 | 9 | 18 | 25
  Chloride: Increase to High | 2 | 2 | 7 | 9
  Carbon dioxide content/Bicarbonate: number analyzed (Participants) | 7 | 8 | 24 | 18
  Carbon dioxide content/Bicarbonate: Decrease Low | 3 | 5 | 12 | 8
  Carbon dioxide content/Bicarbonate: Increase to High | 4 | 3 | 12 | 10
  C-Reactive protein: number analyzed (Participants) | 2 | 0 | 3 | 3
  C-Reactive protein: Decrease Low | 0 | 0 | 0 | 0
  C-Reactive protein: Increase to High | 2 | 0 | 3 | 3
  Creatinine Clearance: number analyzed (Participants) | 7 | 6 | 18 | 11
  Creatinine Clearance: Decrease Low | 5 | 5 | 7 | 7
  Creatinine Clearance: Increase to High | 2 | 1 | 11 | 4
  High Density Lipids cholesterol: number analyzed (Participants) | 0 | 0 | 1 | 0
  High Density Lipids cholesterol: Decrease Low | 0 | 0 | 1 | 0
  High Density Lipids cholesterol: Increase to High | 0 | 0 | 0 | 0
  Lactate Dehydrogenase: number analyzed (Participants) | 9 | 10 | 21 | 24
  Lactate Dehydrogenase: Decrease Low | 2 | 3 | 1 | 4
  Lactate Dehydrogenase: Increase to High | 7 | 7 | 20 | 20
  Low Density Lipids cholesterol: number analyzed (Participants) | 0 | 0 | 1 | 0
  Low Density Lipids cholesterol: Decrease Low | 0 | 0 | 0 | 0
  Low Density Lipids cholesterol: Increase to High | 0 | 0 | 1 | 0
  Total Protein: number analyzed (Participants) | 7 | 8 | 23 | 22
  Total Protein: Decrease Low | 5 | 7 | 17 | 15
  Total Protein: Increase to High | 2 | 1 | 6 | 7
  Troponin I: number analyzed (Participants) | 0 | 0 | 1 | 0
  Troponin I: Decrease Low | 0 | 0 | 0 | 0
  Troponin I: Increase to High | 0 | 0 | 1 | 0
  Troponin T: number analyzed (Participants) | 0 | 0 | 0 | 0
  Troponin T: Decrease Low | 0 | 0 | 0 | 0
  Troponin T: Increase to High | 0 | 0 | 0 | 0
  Urea/BUN: number analyzed (Participants) | 6 | 7 | 22 | 18
  Urea/BUN: Decrease Low | 2 | 2 | 10 | 5
  Urea/BUN: Increase to High | 4 | 5 | 12 | 13

28. Primary Outcome: Part D: Number of Participants With Worst-case Hematology Toxicity Grade Change From Baseline
Description: as for outcome 6
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 15 | 41 | 39
Participants
  Hemoglobin (Increased): number analyzed (Participants) | 0 | 0 | 0 | 0
  Hemoglobin (Increased): Increase to Grade 3 | 0 | 0 | 0 | 0
  Hemoglobin (Increased): Increase to Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin (Anemia): number analyzed (Participants) | 1 | 1 | 3 | 1
  Hemoglobin (Anemia): Increase to Grade 3 | 1 | 1 | 3 | 1
  Hemoglobin (Anemia): Increase to Grade 4 | 0 | 0 | 0 | 0
  Lymphocytes (Increased): number analyzed (Participants) | 0 | 0 | 0 | 0
  Lymphocytes (Increased): Increase to Grade 3 | 0 | 0 | 0 | 0
  Lymphocytes (Increased): Increase to Grade 4 | 0 | 0 | 0 | 0
  Lymphocytes (Decreased): number analyzed (Participants) | 1 | 4 | 12 | 12
  Lymphocytes (Decreased): Increase to Grade 3 | 1 | 3 | 11 | 11
  Lymphocytes (Decreased): Increase to Grade 4 | 0 | 1 | 1 | 1
  Total Neutrophils: number analyzed (Participants) | 0 | 1 | 3 | 4
  Total Neutrophils: Increase to Grade 3 | 0 | 1 | 2 | 4
  Total Neutrophils: Increase to Grade 4 | 0 | 0 | 1 | 0
  Platelet count: number analyzed (Participants) | 1 | 0 | 1 | 0
  Platelet count: Increase to Grade 3 | 1 | 0 | 0 | 0
  Platelet count: Increase to Grade 4 | 0 | 0 | 1 | 0
  White Blood Cell count: number analyzed (Participants) | 0 | 0 | 2 | 3
  White Blood Cell count: Increase to Grade 3 | 0 | 0 | 1 | 3
  White Blood Cell count: Increase to Grade 4 | 0 | 0 | 1 | 0

29. Primary Outcome: Part D: Number of Participants With Worst-case Hematology Change From Baseline With Respect to Normal Range
Description: as for outcome 7
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 15 | 41 | 39
Participants
  Basophils: number analyzed (Participants) | 1 | 2 | 10 | 2
  Basophils: Decrease to Low | 0 | 0 | 2 | 0
  Basophils: Increase to High | 1 | 2 | 8 | 2
  Eosinophils: number analyzed (Participants) | 5 | 4 | 9 | 9
  Eosinophils: Decrease to Low | 1 | 2 | 3 | 4
  Eosinophils: Increase to High | 4 | 2 | 6 | 5
  Erythrocyte Sedimentation Rate: number analyzed (Participants) | 0 | 0 | 0 | 1
  Erythrocyte Sedimentation Rate: Decrease to Low | 0 | 0 | 0 | 0
  Erythrocyte Sedimentation Rate: Increase to High | 0 | 0 | 0 | 1
  Hematocrit: number analyzed (Participants) | 5 | 10 | 21 | 20
  Hematocrit: Decrease to Low | 4 | 10 | 19 | 18
  Hematocrit: Increase to High | 1 | 0 | 2 | 2
  Mean Corpuscle Hemoglobin concentration: number analyzed (Participants) | 9 | 7 | 18 | 12
  Mean Corpuscle Hemoglobin concentration: Decrease to Low | 3 | 4 | 10 | 6
  Mean Corpuscle Hemoglobin concentration: Increase to High | 6 | 3 | 8 | 6
  Mean Corpuscle Hemoglobin: number analyzed (Participants) | 2 | 5 | 15 | 9
  Mean Corpuscle Hemoglobin: Decrease to Low | 1 | 4 | 7 | 6
  Mean Corpuscle Hemoglobin: Increase to High | 1 | 1 | 8 | 3
  Mean Corpuscle Volume: number analyzed (Participants) | 4 | 4 | 10 | 11
  Mean Corpuscle Volume: Decrease to Low | 2 | 4 | 5 | 9
  Mean Corpuscle Volume: Increase to High | 2 | 0 | 5 | 2
  Monocytes: number analyzed (Participants) | 11 | 10 | 29 | 25
  Monocytes: Decrease to Low | 4 | 2 | 12 | 12
  Monocytes: Increase to High | 7 | 8 | 17 | 13
  Red Blood Cell count: number analyzed (Participants) | 5 | 8 | 31 | 18
  Red Blood Cell count: Decrease to Low | 5 | 8 | 26 | 17
  Red Blood Cell count: Increase to High | 0 | 0 | 5 | 1
  Reticulocytes: number analyzed (Participants) | 0 | 0 | 5 | 2
  Reticulocytes: Decrease to Low | 0 | 0 | 3 | 1
  Reticulocytes: Increase to High | 0 | 0 | 2 | 1

30. Primary Outcome: Part D: Number of Participants With the Indicated Worst-case Change From Baseline in Heart Rate and Blood Pressure
Description: Blood pressure were summarized according to National Cancer Institutes (NCI) CTCAE grade, version 4.0. Grade 1, Mild; Grade 2, Moderate; Grade 3 (G3), Severe; Grade 4 (G4), Life-threatening or disabling; Grade 5, Death. Data are presented for only those parameters for which an increase to G3 or G4 occurred.lood pressure measurement included systolic blood pressure (BP, milimeter of mercury [mmHg]) and diastolic BP (DBP). Worst case change from Baseline was calculated as the post-Baseline value minus the Baseline value. Heart Rate is the measure of heartbeats per minute (bpm). Changes in heart rate, either decrease to <60 bpm, change to normal or no change, or increase to >100 bpm are presented
Time Frame: From Baseline (Day 1) until Follow-up visit (up to approximately 7 years)
Population: ATP Population
Measure: Number; unit: Participants
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 15 | 40 | 39
Participants
  Heart rate, Decrease to <60 bpm | 2 | 3 | 12 | 14
  Heart rate, Change to normal or no change | 9 | 8 | 18 | 17
  Heart rate, Increase to >100 bpm | 5 | 5 | 12 | 12
  Systolic BP (mmHg) , increase to G3 or G4 | 3 | 1 | 5 | 6
  Diastolic BP (mmHg), increase to G3 or G4 | 4 | 0 | 2 | 3

31. Secondary Outcome: Part A: Steady State Concentration of Trametinib With Concomitant Administration of Dabrafenib
Description: The steady state plasma concentration (Css) of trametinib with concomitant dabrafenib administration was assessed at Day 15 and Day 16. At steady state the amount of drug administered (in a given time period) is equal to the amount of drug eliminated.
Time Frame: Day 15 and Day 16
Population: PK Population
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part A: Dabrafenib 75 mg + Trametinib 2 mg
Number analyzed (Participants) | 7
ng/mL
  Day 15 | 9.7 [6 to 18]
  Day 16 | 10.2 [6 to 17]

32. Secondary Outcome: Part B: AUC [0-tau] of Dabrafenib (DAB) and Its Metabolite in Combination With Trametinib
Description: Area under the concentration-time curve from time zero (predose) until the last time of quantifiable concentration (AUC [0-tau]) was assessed. Blood samples for PK analysis of dabrafenib and its the metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) were obtained at Day 15 pre-dose and Day 21 pre-dose and at 1, 2, 4, 6, and 8 hours post-dose administration.
Time Frame: Day 15 and Day 21
Population: PK Population. Only those participants who were available at the indicated time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 8 | 12 | 8
ng*hr/mL
  DAB, Day 15 | 2466 [1458 to 4171] | 3539 [1634 to 7666] | 5187 [3737 to 7199] | 4114 [1560 to 10848]
  DAB, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  DAB, Day 21 |  | 4656 [3901 to 5557] | 4528 [3602 to 5692] | 5518 [3732 to 8158]
  GSK2285403, Day 15 | 2120 [1366 to 3290] | 2163 [1267 to 3694] | 3136 [2501 to 3932] | 3180 [1389 to 7283]
  GSK2285403, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2285403, Day 21 |  | 3257 [2162 to 4907] | 2989 [2545 to 3510] | 3632 [2364 to 5581]
  GSK2298683, Day 15 | 37159 [22389 to 61673] | 40634 [30329 to 54441] | 43727 [31486 to 60727] | 68528 [42444 to 110642]
  GSK2298683 , Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2298683 , Day 21 |  | 47911 [30643 to 74909] | 49939 [39219 to 63589] | 59965 [45117 to 79699]
  GSK2167542, Day 15 | 2859 [1568 to 5216] | 2961 [1206 to 7270] | 4156 [2802 to 6165] | 3746 [1992 to 7043]
  GSK2167542, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2167542, Day 21 |  | 3609 [2279 to 5714] | 2995 [1891 to 4743] | 3961 [2361 to 6645]

33. Secondary Outcome: Part B: Pre-dose (Trough) Concentration at the End of the Dosing Interval (Ctau) and Maximum Plasma Concentration (Cmax) of Dabrafenib and Its Metabolite in Combination With Trametinib
Description: Pre-dose (trough) concentration at the end of the dosing interval (Ctau) and maximum plasma concentration (Cmax) were assessed for plasma dabrafenib (DAB) following repeat dosing of DAB administered in combination with trametinib (T). The trough concentration is defined as the plasma level of a pharmaceutical product measured just before the next dose. Blood samples for PK analysis of the metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) of dabrafenib were obtained at Day 15 pre-dose and Day 21 pre-dose and at 1, 2, 4, 6, and 8 hours post-dose administration.
Time Frame: Day 15 and Day 21
Population: PK Population. Only those participants who were available at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 8 | 12 | 8
ng/mL
  DAB Ctau, Day 15 | 59.8 [19.1 to 187] | 44.6 [17.1 to 117] | 115 [27.8 to 472] | 73.7 [10.3 to 528]
  DAB Ctau, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  DAB Ctau, Day 21 |  | 185 [79.7 to 428] | 102 [57.1 to 184] | 79.9 [32.2 to 198]
  DAB Cmax, Day 15 | 640 [390 to 1048] | 906 [221 to 3717] | 1306 [700 to 2437] | 1046 [545 to 2011]
  DAB Cmax, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  DAB Cmax, Day 21 |  | 1263 [863 to 1848] | 1346 [997 to 1817] | 1391 [1002 to 1932]
  GSK2285403 Ctau, Day 15 | 72.9 [25.2 to 211] | 47.8 [20.2 to 113] | 97.9 [32.2 to 297] | 74.4 [15.7 to 353]
  GSK2285403 Ctau, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2285403 Ctau, Day 21 |  | 136 [62.4 to 299] | 92.9 [60.2 to 143] | 82.7 [37.6 to 182]
  GSK2285403 Cmax, Day 15 | 399 [265 to 601] | 418 [146 to 1201] | 597 [300 to 1186] | 630 [411 to 964]
  GSK2285403 Cmax, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2285403 Cmax, Day 21 |  | 775 [441 to 1364] | 668 [507 to 882] | 722 [502 to 1039]
  GSK2298683 Ctau, Day 15 | 2345 [1237 to 4447] | 2360 [1134 to 4911] | 2792 [2069 to 3768] | 4372 [2589 to 7384]
  GSK2298683 Ctau, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2298683 Ctau, Day 21 |  | 2920 [1674 to 5095] | 3221 [2619 to 3962] | 3740 [2564 to 5455]
  GSK2298683 Cmax, Day 15 | 3757 [2385 to 5916] | 4545 [3817 to 5411] | 4636 [3258 to 6598] | 7098 [4914 to 10254]
  GSK2298683 Cmax, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2298683 Cmax, Day 21 |  | 5301 [3392 to 8286] | 5416 [4163 to 7048] | 6257 [4937 to 7931]
  GSK2167542 Ctau, Day 15 | 257 [140 to 473] | 249 [79.4 to 782] | 331 [185 to 590] | 318 [260 to 389]
  GSK2167542 Ctau, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2167542 Ctau, Day 21 |  | 196 [90.8 to 425] | 248 [140 to 439] | 369 [191 to 714]
  GSK2167542 Cmax, Day 15 | 300 [157 to 572] | 355 [114 to 1108] | 523 [251 to 1091] | 460 [190 to 1113]
  GSK2167542 Cmax, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2167542 Cmax, Day 21 |  | 543 [298 to 989] | 373 [248 to 562] | 430 [226 to 818]

34. Secondary Outcome: Part B: Tmax of Dabrafenib and Its Metabolite in Combination With Trametinib
Description: The tmax is defined as the time of occurenceof Cmax. Tha tmax was assessed for plasma dabrafenib (DAB) following repeat dosing of dabrafenib 75 and 150 mg BID administered in combination with trametinib. Blood samples for PK analysis of the metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) of dabrafenib were obtained at Day 15 pre-dose and Day 21 pre-dose and at 1, 2, 4, 6, and 8 hours post-dose administration.
Time Frame: Day 15 and Day 21
Population: PK Population. Only those participants who were available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 8 | 12 | 8
Hours
  DAB Day 15 | 2.00 [1.03 to 2.00] | 2.00 [1.03 to 6.00] | 2.00 [1.00 to 2.10] | 1.50 [1.00 to 2.00]
  DAB Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  DAB Day 21 |  | 1.54 [1.00 to 2.00] | 1.53 [1.00 to 2.03] | 2.04 [1.00 to 4.03]
  GSK2285403 Day 15 | 2.00 [2.00 to 2.03] | 2.00 [1.03 to 8.00] | 2.00 [2.00 to 4.03] | 2.00 [2.00 to 2.00]
  GSK2285403 Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2285403 Day 21 |  | 1.97 [0.00 to 2.00] | 2.00 [1.00 to 2.03] | 2.07 [1.00 to 6.00]
  GSK2298683 Day 15 | 6.00 [4.00 to 8.00] | 4.96 [0.00 to 6.30] | 4.17 [1.00 to 8.02] | 4.10 [4.00 to 8.00]
  GSK2298683 Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2298683 Day 21 |  | 4.00 [1.00 to 6.00] | 4.00 [1.00 to 6.00] | 4.02 [2.00 to 8.07]
  GSK2167542 Day 15 | 0.00 [0.00 to 4.17] | 2.94 [0.00 to 8.00] | 4.17 [1.00 to 8.02] | 1.52 [0.00 to 2.00]
  GSK2167542 Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  GSK2167542 Day 21 |  | 2.00 [1.00 to 2.32] | 1.01 [0.00 to 8.00] | 1.50 [0.00 to 8.15]

35. Secondary Outcome: Part B (Analyte=GSK1120212): AUC (0-tau) Assessment of Trametinib in Combination With Dabrafenib
Description: AUC (0-tau) is defined as area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration. AUC (0-tau) was assessed for plasma trametinib following repeat dosing of trametinib in combination with dabrafenib. Blood samples for PK analysis of the metabolites of dabrafenib were obtained at Day 15 pre-dose and Day 21 pre-dose and at 1, 2, 4, 6, and 8 hours post-dose administration.
Time Frame: Day 15 and Day 21
Population: PK Population. Only those participants who were available at the indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 8 | 12 | 8
ng*hr/mL
  Day 15 | 169 [113 to 252] | 147 [101 to 212] | 217 [139 to 338] | 394 [229 to 679]
  Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  Day 21 |  | 169 [146 to 194] | 269 [238 to 304] | 351 [284 to 432]

36. Secondary Outcome: Part B (Analyte=GSK1120212): Ctau and Cmax Assessments of Trametinib in Combination With Dabrafenib
Description: Pre-dose (trough) concentration at the end of the dosing interval (Ctau) and maximum plasma concentration (Cmax) were assessed for plasma trametinib following repeat dosing of trametinib in combination with dabrafenib. Blood samples for PK analysis of the metabolites of dabrafenib were obtained at Day 15 pre-dose or Day 21 pre-dose and at 1, 2, 4, 6, and 8 hours post-dose administration.
Time Frame: Day 15 and Day 21
Population: PK Population. Only those participants who were available at the indicated time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 8 | 12 | 8
ng/mL
  Ctau, Day 15 | 5.56 [3.74 to 8.28] | 5.05 [3.81 to 6.69] | 7.62 [5.38 to 10.8] | 12.4 [6.50 to 23.6]
  Ctau, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  Ctau, Day 21 |  | 5.57 [4.80 to 6.45] | 8.51 [7.65 to 9.48] | 10.8 [8.75 to 13.3]
  Cmax, Day 15 | 10.2 [7.18 to 14.4] | 8.08 [5.06 to 12.9] | 11.5 [6.16 to 21.5] | 22.4 [14.0 to 35.6]
  Cmax, Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  Cmax, Day 21 |  | 10.2 [8.50 to 12.1] | 18.0 [14.9 to 21.7] | 22.6 [18.1 to 28.2]

37. Secondary Outcome: Part B (Analyte=GSK1120212): Tmax Assessment of Trametinib in Combination With Dabrafenib
Description: The tmax is defined as the time of occurrence of Cmax. The PK parameter for tmax was assessed for plasma trametinib following repeat dosing of trametinib in combination with dabrafenib. Blood samples for PK analysis of the metabolites of dabrafenib were obtained at Day 15 pre-dose or Day 21 pre-dose and at 1, 2, 4, 6, and 8 hours post-dose administration.
Time Frame: Day 15 and Day 21
Population: PK Population. Only those participants who were available at the indicated time point were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 8 | 12 | 8
Hours
  Day 15 | 2.00 [1.03 to 4.00] | 2.00 [1.00 to 8.00] | 2.00 [1.00 to 8.00] | 1.52 [1.00 to 2.00]
  Day 21: number analyzed (Participants) | 0 | 8 | 12 | 8
  Day 21 |  | 2.00 [0.93 to 8.00] | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 8.15]

38. Secondary Outcome: Part B: Number of Participants With BRAFi-naïve Mutant Metastatic Melanoma With the Best Overall Response as Assessed by Investigator
Description: Best overall response is defined as complete response (CR: the disappearance of all target lesions. Any pathological lymph nodes must be <10 milimeter [mm] in the short axis.) or partial reponse (PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). Participants with unknown or missing response were considered as non-responders. To be assigned a status of PR or CR, a confirmatory disease assessment should have been performed no less than 28 days after the criteria for response were first met. Response was evaluated by an investigator as per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. BRAFi-naïve participants were those with BRAF-mutation-positive melanoma who had not received prior therapy with a BRAF inhibitor.
Time Frame: From the first dose of study medication to the first documented evidence of a confirmed complete response or partial response (up to approximately 8 years)
Population: All Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 22 | 25 | 24
Participants
  CR | 0 | 4 | 3 | 4
  PR | 4 | 10 | 8 | 11

39. Secondary Outcome: Part B: Duration of Response as Assessed by the Investigator in Participants With BRAFi-naïve Mutant Metastatic Melanoma
Description: Duration of response for participants with either a CR (the disappearance of all target lesions. Any pathological lymph nodes must be <10 mm in the short axis.) or PR (at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]) is defined as the time from the first documented evidence of a PR or CR until the first documented sign of disease progression (PD) or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. BRAFi-naïve participants were those with BRAF-mutation-positive melanoma who had not received prior therapy with a BRAF inhibitor.
Time Frame: First documented evidence of PR or CR until the earlier of date of disease progression or date of death due to any cause (up to approximately 8 years)
Population: All Treated Population. Only those participants who had a CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 22 | 25 | 24
Months | 12.4 [3.7 to NA] — NA: Not estimable due to insufficient number of participants with events | 8.4 [3.9 to 27.4] | 12.6 [5.1 to NA] — NA: Not estimable due to insufficient number of participants with events | 16.9 [7.4 to NA] — NA: Not estimable due to insufficient number of participants with events

40. Secondary Outcome: Part B: Progression-free Survival (PFS) as Assessed by the Investigator in Participants With BRAFi-naïve Mutant Metastatic Melanoma
Description: PFS is defined as the interval between the first dose of study medication and the earliest date of PD or death due to any cause. PD was based on radiographic or photographic evidence, and assessments were made by the investigator according to RECIST, version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm. BRAFi-naïve were the participants with BRAF-mutation positive melanoma who had not received prior therapy with a BRAF-inhibitor..
Time Frame: From the date of first dose to the earliest date of disease progression (PD) or death due to any cause (up to approximately 8 years)
Population: All Treated Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 22 | 25 | 24
Months | 8.7 [3.4 to NA] — NA: Not estimable due to insufficient number of participants with events | 8.2 [4.3 to 11.0] | 5.4 [3.5 to 12.8] | 10.8 [3.6 to 18.6]

41. Secondary Outcome: Part B: Overall Survival (OS) in BRAFi Naïve Melanoma Participants
Description: OS is defined as the interval of time between the first dose of study medication until the date of death due to any cause. For the participants who did not die, overall survival was censored at the date of last contact.
Time Frame: From the date of first dose until date of death due to any cause (up to approximately 8 years)
Population: All Treated Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 6 | 22 | 25 | 24
Months | 17.4 [8.0 to NA] — NA: Not estimable due to insufficient number of participants with events | 23.5 [12.9 to 33.7] | 13.3 [6.3 to 23.4] | 41.5 [12.9 to NA] — NA: Not estimable due to insufficient number of participants with events

42. Secondary Outcome: Part B: Pre- and Post-dose H-scores for Individual Participants
Description: p-ERK and p-AKT, biomarkers in tumor biopsies, were assessed for participants with BRAF mutant colorectal cancer. The H-score, which is a composite score that comprises intensity and percentage of staining, is a method of assessing the amount of protein or phospho-protein present in a biopsy sample. The score is obtained by the formula: (3 * percentage of strongly staining nuclei) + (2 * percentage of moderately staining nuclei) + (percentage of weakly staining nuclei). The H-score ranges from 0 to 300, with a score of 0 representing the absence of any of the target protein and an H-score of 300 representing maximum staining and intensity of the target protein.
Time Frame: Screening and at disease progression (up to approximately 8 years)
Population: Biomarker Population: participants with H-score data for pre- and post-biopsy pairs
Measure: Number; unit: scores on a scale
Groups:
- Part B: Dabrafenib + Trametinib: Melanoma BRAF-positive participants who did not receive prior treatment with BRAF inhibitors received dabrafenib (75 mg or 150 mg) gelatin capsules BID and trametinib (1 mg, 1.5 mg, or 2 mg) tablets QD as continuous daily dosing. Dose escalation decisions were made based on all available pharmacokinetic (PK), safety, and other data from the first 4 evaluable participants, and additional participants were enrolled based on dose-limiting toxicities (DLTs) occurring during the first 3 weeks of treatment.
Arm/Group | Part B: Dabrafenib + Trametinib
Number analyzed (Participants) | 10
scores on a scale
  p-ERK: Participant 1, pre-dose score | 135
  p-ERK: Participant 1, post-dose score | 109
  p-ERK: Participant 2, pre-dose score | 193
  p-ERK: Participant 2, post-dose score | 138
  p-ERK: Participant 3, pre-dose score | 148
  p-ERK: Participant 3, post-dose score | 65
  p-ERK: Participant 4, pre-dose score | 80
  p-ERK: Participant 4, post-dose score | 20
  p-ERK: Participant 5, pre-dose score | 130
  p-ERK: Participant 5, post-dose score | 99
  p-ERK: Participant 6, pre-dose score | 68
  p-ERK: Participant 6, post-dose score | 7
  p-ERK: Participant 7, pre-dose score | 128
  p-ERK: Participant 7, post-dose score | 81
  p-ERK: Participant 8, pre-dose score | 196
  p-ERK: Participant 8, post-dose score | 75
  p-ERK: Participant 9, pre-dose score | 164
  p-ERK: Participant 9, post-dose score | 109
  p-ERK: Participant 10, pre-dose score | 239
  p-ERK: Participant 10, post-dose score | 78
  p-AKT: Participant 1, pre-dose score | 130
  p-AKT, Participant 1, post-dose score | 180
  p-AKT: Participant 2, pre-dose score | 76
  p-AKT, Participant 2, post-dose score | 50
  p-AKT: Participant 3, pre-dose score | 192
  p-AKT, Participant 3, post-dose score | 277
  p-AKT: Participant 4, pre-dose score | 25
  p-AKT, Participant 4, post-dose score | 135
  p-AKT: Participant 5, pre-dose score | 55
  p-AKT, Participant 5, post-dose score | 2
  p-AKT: Participant 6, pre-dose score | 145
  p-AKT, Participant 6, post-dose score | 20
  p-AKT: Participant 7, pre-dose score | 22
  p-AKT, Participant 7, post-dose score | 7
  p-AKT: Participant 8, pre-dose score | 183
  p-AKT, Participant 8, post-dose score | 123
  p-AKT: Participant 9, pre-dose score | 278
  p-AKT, Participant 9, post-dose score | 289
  p-AKT: Participant 10, pre-dose score | 73
  p-AKT, Participant 10, post-dose score | 0

43. Secondary Outcome: Part C (Randomized): Overall Survival (OS)
Description: OS is defined as the interval of time between the date of randomization until the date of death due to any cause. For the participants who did not die, overall survival was censored at the date of last contact. When calculating overall survival, deaths following crossover were included.
Time Frame: From the date of randomization until date of death due to any cause (up to approximately 7 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 54 | 54 | 54
Months | 20.2 [14.0 to 27.1] | 18.7 [13.7 to 35.3] | 25.0 [17.5 to 36.5]

44. Secondary Outcome: Part C: Plasma Concentrations of Dabrafenib and Its Metabolites
Description: Plasma concentrations of dabrafenib and its metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) were assesed following daily dose of dabrafenib and trametinib.
Time Frame: Day 15, Week 8, Week 16, Week 24, Week 32, Week 40, Week 48, and Week 56
Population: PK Population. Only those participants who were available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 49 | 53 | 50
ng/mL
  Day 15, GSK2118436 | 59.3 [9 to 2420] | 68.2 [0 to 1555] | 66.3 [7 to 1804]
  Week 8, GSK2118436 | 45.6 [3 to 1841] | 69.8 [0 to 946] | 50.5 [0 to 1696]
  Week 16, GSK2118436 | 84.4 [0 to 1865] | 66.7 [0 to 1774] | 82.9 [2 to 3033]
  Week 24, GSK2118436 | 66.3 [4 to 594] | 66.2 [1 to 2684] | 93.3 [7 to 741]
  Week 32, GSK2118436 | 40.6 [1 to 500] | 57.1 [0 to 1424] | 66.4 [0 to 2042]
  Week 40, GSK2118436 | 229 [5 to 714] | 97.6 [19 to 2597] | 150.9 [0 to 1624]
  Week 48, GSK2118436 | 44.7 [13 to 132] | 105.6 [0 to 1322] | 107.7 [3 to 806]
  Week 56, GSK2118436 | 46.4 [25 to 68] | 44.5 [0 to 6646] | 193.8 [3 to 413]
  Day 15, GSK2285403 | 92.7 [14 to 1337] | 71.8 [2 to 1220] | 90.5 [10 to 995]
  Week 8, GSK2285403 | 65.2 [3 to 2041] | 80.4 [0 to 769] | 90.6 [0 to 757]
  Week 16, GSK2285403 | 113.4 [0 to 2090] | 81.9 [0 to 995] | 114.7 [3 to 2563]
  Week 24, GSK2285403 | 95.0 [4 to 616] | 88.1 [0 to 1689] | 130.2 [9 to 529]
  Week 32, GSK2285403 | 62.5 [3 to 890] | 86.7 [0 to 808] | 87.4 [0 to 973]
  Week 40, GSK2285403 | 263.8 [7 to 693] | 143.5 [16 to 870] | 136.2 [0 to 1665]
  Week 48, GSK2285403 | 43.3 [32 to 241] | 93.6 [0 to 898] | 146.4 [2 to 418]
  Week 56, GSK2285403 | 48.3 [45 to 51] | 92.9 [0 to 1841] | 141.5 [7 to 755]
  Day 15, GSK2298683 | 3493 [1381 to 16820] | 3043.3 [199 to 8562] | 3145.8 [428 to 16240]
  Week 8, GSK2298683 | 3149.7 [238 to 13330] | 3238.4 [20 to 7686] | 3010 [31 to 13130]
  Week 16, GSK2298683 | 3497.9 [21 to 9952] | 2946.1 [0 to 8782] | 2756.5 [44 to 14004]
  Week 24, GSK2298683 | 2876.5 [500 to 8635] | 3365.4 [25 to 7482] | 3193.7 [133 to 6531]
  Week 32, GSK2298683 | 2699.9 [447 to 14341] | 3267.1 [0 to 9278] | 3046.8 [50 to 9077]
  Week 40, GSK2298683 | 4410.6 [1023 to 14258] | 3694.7 [1900 to 7663] | 3492.8 [0 to 12550]
  Week 48, GSK2298683 | 3554.9 [1889 to 7148] | 4146.9 [0 to 8351] | 3936.1 [464 to 12239]
  Week 56, GSK2298683 | 2032.2 [1102 to 2963] | 3843.5 [374 to 6866] | 2904.9 [1305 to 4673]
  Day 15, GSK2167542 | 247.9 [95 to 955] | 288 [49 to 1164] | 289.3 [72 to 1140]
  Week 8, GSK2167542 | 239.5 [19 to 1092] | 275.2 [3 to 983] | 262.4 [0 to 9876]
  Week 16, GSK2167542 | 244 [1 to 772] | 204.4 [0 to 922] | 243.8 [3 to 1049]
  Week 24, GSK2167542 | 225.6 [48 to 899] | 247.2 [4 to 990] | 254.6 [3 to 846]
  Week 32, GSK2167542 | 171 [19 to 544] | 255.4 [0 to 698] | 289.3 [2 to 962]
  Week 40, GSK2167542 | 222.2 [95 to 639] | 249.3 [55 to 674] | 268.9 [0 to 910]
  Week 48, GSK2167542 | 204.5 [145 to 286] | 232 [0 to 915] | 260.9 [81 to 886]
  Week 56, GSK2167542 | 171.8 [116 to 228] | 250 [28 to 851] | 462.1 [107 to 663]

45. Secondary Outcome: Part C: Plasma Concentrations of Trametinib
Description: Plasma concentrations of trametinib was assessed following daily dose of dabrafenib and trametinib.
Time Frame: Day 15, Week 8, Week 16, Week 24, Week 32, Week 40, Week 48, and Week 56
Population: PK Population. Only those participants who were available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Dabrafenib 150 mg + Trametinib 1 mg | Part C: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 59 | 53 | 50
ng/mL
  Day 15 | 0 [0 to 0] | 5.86 [3.4 to 11.3] | 9.35 [4.8 to 26.00]
  Week 8 | 0 [0 to 13.9] | 6.70 [2.0 to 9.6] | 10.3 [0 to 25.8]
  Week 16 | 0 [0 to 9.8] | 6.99 [0 to 20.7] | 9.87 [1.1 to 25.4]
  Week 24 | 0 [0 to 19.7] | 5.99 [0 to 11.2] | 9.54 [0.5 to 27.4]
  Week 32 | 0 [0 to 0] | 5.77 [0.7 to 11.6] | 9.74 [0 to 51.5]
  Week 40 | 0 [0 to 0] | 7.11 [2.2 to 16.7] | 10.1 [0 to 26.4]
  Week 48 | 0 [0 to 0] | 5.62 [0 to 14.3] | 10.3 [0 to 35.6]
  Week 56 | 0 [0 to 0] | 9.90 [3.4 to 16.9] | 8.60 [0 to 15.4]

46. Secondary Outcome: Part C: Oral Clearance (CL/F) of Dabrafenib and Trametinib
Description: Oral clearance (CL/F) of dabrafenib and trametinib were assessed using a population approach. Oral clearance (CL/F) is defined as the apparent volume of plasma in the vascular compartment cleared of drug per unit time by the processes of metabolism and excretion. For dabrafenib, population CL/F is defined as inducible and non-inducible CL/F. As dabrafenib induces its own metabolism, total oral clearance at steady state includes a non-induced (Day 1) component and an induced component, as estimated by a population PK model.
Time Frame: Day 15, Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: PK Population
Measure: Mean (95% Confidence Interval); unit: Liters per hour (L/hr)
Groups:
- Part C: Trametinib: Participants received Trametinib 1 mg or 2 mg tablets QD.
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Trametinib
Number analyzed (Participants) | 53 | 109
Liters per hour (L/hr)
  Non-inducible | 19.4 [17.6 to 21.2] | 5.07 [4.83 to 5.31]
  Inducible: number analyzed (Participants) | 53 | 0
  Inducible | 20.0 [19.2 to 20.8] |

47. Secondary Outcome: Part C: Oral Volume of Distribution (V/F) of Dabrafenib and Trametinib
Description: Oral volume of distribution (V/F) of dabrafenib and trametinib were assessed using a population approach. Oral volume of distribution (V/F) is defined as the apparent volume of distribution in the central compartment.
Time Frame: Day 15, Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48
Population: PK Population
Measure: Mean (95% Confidence Interval); unit: Liters (L)
Arm/Group | Part C: Dabrafenib 150 mg | Part C: Trametinib
Number analyzed (Participants) | 53 | 109
Liters (L) | 80.8 [73.9 to 87.7] | 184 [158 to 210]

48. Secondary Outcome: Part D: Cmax of Dabrafenib Metabolites
Description: The maximum concentration (Cmax) of dabrafenib metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) after single and repeat doses of DAB alone and in combination with trametinib was measured at Day 1 and Day 21.
Time Frame: Day 1: pre-dose, and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 24 hours post dose. Day 21: pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, and 10 hours post-dose
Population: PK Population. Only participants who were available at the indicated timepoints were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15
ng/mL
  GSK2285403, Day 1 | 525 [429 to 643] | 1055 [705 to 1579] | 597 [474 to 752] | 1363 [300 to 2066]
  GSK2285403, Day 21 | 596 [501 to 709] | 1203 [906 to 1599] | 696 [551 to 880] | 1120 [725 to 1730]
  GSK2298683, Day 1 | 1475 [1249 to 1741] | 2268 [1595 to 3223] | 1478 [1197 to 1824] | 2551 [1756 to 3707]
  GSK2298683, Day 21 | 3637 [3119 to 4242] | 6743 [5133 to 8859] | 4158 [3136 to 5514] | 6319 [4725 to 8450]
  GSK2167542, Day 1 | 50.1 [30 to 84] | 68.6 [36 to 129] | 61.2 [41 to 91] | 86.3 [48 to 155]
  GSK2167542, Day 21 | 210 [154 to 285] | 355 [268 to 470] | 289 [201 to 416] | 440 [303 to 637]

49. Secondary Outcome: Part D: Tmax of Dabrafenib Metabolites
Description: The time to Cmax (tmax) of DAB metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) after single and repeat doses of DAB alone and in combination with trametinib was measuered at Day 1 and Day 21.
Time Frame: as for outcome 48
Population: PK Population. Only participants who were available at the indicated timepoints were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15
Hours
  GSK2285403, Day 1 | 3.00 [1.50 to 4.00] | 3.51 [2.00 to 6.18] | 3.00 [2.00 to 6.02] | 2.07 [1.50 to 10.00]
  GSK2285403, Day 21 | 2.00 [1.50 to 3.00] | 2.00 [1.42 to 3.00] | 2.00 [1.47 to 4.00] | 2.00 [1.00 to 3.98]
  GSK2298683, Day 1 | 10.0 [5.98 to 10.1] | 8.93 [4.00 to 24.0] | 10.0 [6.00 to 24.0] | 8.00 [4.07 to 24.0]
  GSK2298683, Day 21 | 5.00 [3.00 to 8.00] | 4.00 [3.00 to 6.00] | 5.98 [2.00 to 10.00] | 4.00 [3.00 to 6.08]
  GSK2167542, Day 1 | 24.0 [8.00 to 24.1] | 24.0 [6.00 to 24.6] | 24.0 [23.5 to 25.0] | 24.0 [10.0 to 24.3]
  GSK2167542, Day 21 | 0.75 [0 to 10.0] | 2.00 [0.50 to 10.0] | 2.00 [1.00 to 10.00] | 1.75 [0 to 9.92]

50. Secondary Outcome: Part D: Area Under the Concentration-time Curve (AUC) of Dabrafenib Metabolites
Description: Area under the concentration-time curve (AUC) from pre-dose to dosing interval (AUC[0-tau]), from pre-dose to the last time of quantifable concentration (AUC[0-tau]), and from pre-dose extrapolated to infinity (AUC[0-inf]) of DAB metabolites hydroxy-dabrafenib (GSK2285403), carboxy-dabrafenib (GSK2298683) and desmethyl-dabrafenib (GSK2167542) after single and repeat doses of DAB alone and in combination with trametinib was measured at Day 1 and Day 21.
Time Frame: as for outcome 48
Population: PK Population. Only participants who were available at the indicated timepoints were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 15 | 14 | 15 | 15
ng*hr/mL
  GSK2285403, AUC(0-tau), Day 1 | 3134 [2533 to 3877] | 5950 [4045 to 8753] | 3694 [2903 to 4700] | 6524 [4520 to 9416]
  GSK2285403, AUC(0-inf), Day 1 | 3963 [3147 to 4990] | 7415 [4991 to 11015] | 5026 [3934 to 6422] | 7907 [5434 to 11506]
  GSK2285403, AUC (0-tau), Day 21 | 2568 [2099 to 3143] | 4262 [3007 to 6040] | 2919 [2296 to 3711] | 4216 [2986 to 5951]
  GSK2298683, AUC, (0-tau), Day 1 | 10396 [8388 to 12885] | 15952 [10532 to 24160] | 9575 [7143 to 12835] | 20935 [12430 to 35259]
  GSK2298683, AUC (0-t), Day 1 | 20047 [15384 to 26125] | 35206 [24970 to 49639] | 22692 [18398 to 27988] | 31666 [18474 to 54277]
  GSK2298683, AUC (0-tau), Day 21 | 34283 [29189 to 40266] | 59340 [44595 to 78960] | 39672 [29504 to 53343] | 52712 [40084 to 69318]
  GSK2167542, AUC(0-tau), Day 1 | 132 [79 to 219] | 190 [101 to 356] | 88.8 [56 to 139] | 354 [228 to 549]
  GSK2167542, AUC(0-t) Day 1 | 500 [271 to 925] | 737 [385 to 1410] | 614 [415 to 906] | 1316 [824 to 2103]
  GSK2167542, AUC(0-tau), Day 21 | 1775 [1225 to 2570] | 2707 [2106 to 3481] | 2508 [1793 to 3507] | 3632 [2529 to 5216]

51. Secondary Outcome: Part D: Cmax Assessment of Trametinib
Description: Cmax of trametinib after single and repeat dose in combination with DAB was observed at Day 1 and Day 21. Blood samples for PK analysis of dabrafenib were obtained at pre-dose Day 1 and Day 21 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours (Day 1 only) post-dose administration. From the plasma concentration-time curve, the PK parameter tmax was determined by standard non-compartmental analysis using WinNonlin.Participants receiving DAB 75 mg to DAB 75 mg + Trametinib 2 mg and those receiving DAB 150 mg to DAB 150 mg + Trametinib 2 mg did not receive Trametinib until Day 29; therefore, Cmax was not analyzed in these participants at Days 1 and 21.
Time Frame: as for outcome 48
Population: PK Population. Only participants who were available at the indicated timepoints were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 0 | 0 | 15 | 14
ng/mL
  Day 1 |  |  | 6.8 [5 to 10] | 6.6 [4 to 10]
  Day 21 |  |  | 24.1 [20 to 29] | 22.6 [20 to 26]

52. Secondary Outcome: Part D: Tmax Assessment of Trametinib
Description: The tmax of trametinib after single and repeat dose in combination with dabrafenib (DAB) was observed at Day 1 and Day 21. Blood samples for PK analysis of dabrafenib were obtained at pre-dose Day 1 and Day 21 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours (Day 1 only) post-dose administration. From the plasma concentration-time curve, the PK parameter tmax was determined by standard non-compartmental analysis using WinNonlin.Participants receiving DAB 75 mg to DAB 75 mg + Trametinib 2 mg and those receiving DAB 150 mg to DAB 150 mg + Trametinib 2 mg did not receive Trametinib until Day 29; therefore, tmax was not analyzed in these participants at Days 1 and 21.
Time Frame: as for outcome 48
Population: PK Population. Only participants who were available at the indicated timepoints were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 0 | 0 | 15 | 14
Hours
  Day 1 |  |  | 2.00 [1.00 to 3.00] | 1.50 [1.00 to 8.00]
  Day 21 |  |  | 2.00 [1.00 to 4.00] | 2.00 [1.50 to 3.98]

53. Secondary Outcome: Part D: Area Under the Concentration-time Curve Assessment of Trametinib
Description: AUC(0-tau) after single and repeat dose of teametinib alone and in combination with dabrafenib was observed at Day 1 and Day 21. Blood samples for PK analysis of dabrafenib were obtained at pre-dose Day 1 and Day 21 pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours (Day 1 only) post-dose administration. From the plasma concentration-time curve, the PK parameter tmax was determined by standard non-compartmental analysis using WinNonlin.Participants receiving DAB 75 mg to DAB 75 mg + Trametinib 2 mg and those receiving DAB 150 mg to DAB 150 mg + Trametinib 2 mg did not receive Trametinib until Day 29; therefore, AUC(0-tau) was not analyzed in these participants at Days 1 and 21.
Time Frame: as for outcome 48
Population: PK Population. Only participants who were available at the indicated timepoints were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 0 | 0 | 15 | 14
ng*h/mL
  Day 1 |  |  | 53.4 [40 to 72] | 50.7 [39 to 66]
  Day 21 |  |  | 366 [305 to 439] | 356 [318 to 400]

54. Secondary Outcome: Part D: Number of Participants With the Best Overall Response as Assessed by the Investigator in Participants
Description: Best overall response is defined as complete response (CR: the disappearance of all target lesions. Any pathological lymph nodes must be <10 milimeter [mm] in the short axis.) or partial reponse (PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters [e.g., percent change from Baseline]). To be assigned a status of PR or CR, a confirmatory disease assessment should be performed no less than 28 days after the criteria for response are first met. Response was evaluated by an investigator as per Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
Time Frame: From the date of first dose of study medication to the first documented evidence of a confirmed complete response or partial response (up to approximately 7 years)
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 12 | 16 | 43 | 39
Participants
  CR | 0 | 2 | 5 | 7
  PR | 8 | 10 | 28 | 21

55. Secondary Outcome: Part D: Duration of Response as Assessed by the Investigator
Description: as for outcome 15
Time Frame: First documented evidence of PR or CR until the earlier of date of disease progression or date of death due to any cause (up to approximately 7 years)
Population: ITT Population. Only those participants who had CR or PR were considered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 12 | 16 | 43 | 39
Months | 8.2 [3.5 to 14.8] | 10.1 [5.6 to NA] — NA: Not estimable due to insufficient number of participants with events | 5.9 [3.7 to 9.0] | 14.3 [8.8 to 67.8]

56. Secondary Outcome: Part D: Progression-free Survival (PFS) as Assessed by the Investigator
Description: PFS is defined as the interval between the date of randomization and the earliest date of PD or death due to any cause. PD was based on radiographic or photographic evidence, and assessments were made by the investigator according to RECIST, version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: as for outcome 12
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 12 | 16 | 43 | 39
Months | 7.9 [3.4 to 11.4] | 9.3 [3.7 to 28.6] | 7.4 [5.6 to 10.7] | 11.1 [7.0 to 28.5]

57. Secondary Outcome: Part D: Overall Survival (OS)
Description: OS is defined as the interval of time between the date of randomization until the date of death due to any cause. For the participants who did not die, overall survival was censored at the date of last contact.
Time Frame: From the date of first dose until date of death due to any cause (up to approximately 7 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
Number analyzed (Participants) | 12 | 16 | 43 | 39
Months | 19.5 [12.4 to 28.0] | 15.5 [10.4 to 60.0] | 15.3 [13.0 to 37.2] | 40.3 [15.7 to 69.6]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 90 months.
Arm/Group | Part A: Dabrafenib 75 mg + Trametinib 2 mg | Part B: Dabrafenib 75 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1 mg | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg | Part B: Dabrafenib 150 mg + Trametinib 2 mg | Part C (Randomized): Dabrafenib 150 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg | Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg | Part D: Dabrafenib 75 mg + Trametinib 2 mg | Part D: Dabrafenib 150 mg + Trametinib 2 mg
All-Cause Mortality (participants affected / at risk) | 2/8 | 0/6 | 1/23 | 6/27 | 12/94 | 1/53 | 4/54 | 7/55 | 7/45 | 1/15 | 4/15 | 7/41 | 2/39
Serious Adverse Events (participants affected / at risk) | 5/8 | 1/6 | 15/23 | 14/27 | 55/94 | 15/53 | 24/54 | 39/55 | 24/45 | 8/15 | 11/15 | 29/41 | 30/39
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 23/23 | 27/27 | 91/94 | 53/53 | 53/54 | 55/55 | 44/45 | 15/15 | 15/15 | 41/41 | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Dabrafenib 75 mg + Trametinib 2 mg (N=8) | Part B: Dabrafenib 75 mg + Trametinib 1 mg (N=6) | Part B: Dabrafenib 150 mg + Trametinib 1 mg (N=23) | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg (N=27) | Part B: Dabrafenib 150 mg + Trametinib 2 mg (N=94) | Part C (Randomized): Dabrafenib 150 mg (N=53) | Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg (N=54) | Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg (N=55) | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg (N=45) | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg (N=15) | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg (N=15) | Part D: Dabrafenib 75 mg + Trametinib 2 mg (N=41) | Part D: Dabrafenib 150 mg + Trametinib 2 mg (N=39)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Addison's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 3 | 0 | 3 | 1 | 2 | 0 | 0 | 2 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 4 | 0 | 1 | 0 | 0 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 3 | 2 | 18 | 1 | 7 | 12 | 5 | 6 | 5 | 14 | 15
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hernia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 6 | 6 | 25 | 1 | 10 | 16 | 7 | 6 | 6 | 16 | 16
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder enlargement (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to immunoglobulin therapy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 5
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pelvic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 1 | 2
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Ejection fraction (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 8 | 0 | 3 | 4 | 5 | 1 | 0 | 3 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 4 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 3
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 3
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 3 | 2 | 6 | 0 | 2 | 4 | 0 | 1 | 2 | 4
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cervical cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Focal dyscognitive seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Sensory ganglionitis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 1 | 0 | 1 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Granulomatous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 3 | 7 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Dabrafenib 75 mg + Trametinib 2 mg (N=8) | Part B: Dabrafenib 75 mg + Trametinib 1 mg (N=6) | Part B: Dabrafenib 150 mg + Trametinib 1 mg (N=23) | Part B: Dabrafenib 150 mg + Trametinib 1.5 mg (N=27) | Part B: Dabrafenib 150 mg + Trametinib 2 mg (N=94) | Part C (Randomized): Dabrafenib 150 mg (N=53) | Part C (Randomized): Dabrafenib 150 mg + Trametinib 1 mg (N=54) | Part C (Randomized): Dabrafenib 150 mg + Trametinib 2 mg (N=55) | Part C (Crossover): Dabrafenib 150 mg + Trametinib 2 mg (N=45) | Part D: Dabrafenib (DAB) 75 mg to DAB 75 mg + Trametinib 2 mg (N=15) | Part D: Dabrafenib 150 mg to DAB 150 mg + Trametinib 2 mg (N=15) | Part D: Dabrafenib 75 mg + Trametinib 2 mg (N=41) | Part D: Dabrafenib 150 mg + Trametinib 2 mg (N=39)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 3 | 21 | 3 | 10 | 12 | 9 | 0 | 6 | 8 | 8
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 3 | 8 | 2 | 2 | 2 | 3 | 0 | 0 | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 6 | 11 | 1 | 8 | 4 | 2 | 1 | 2 | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3 | 10 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0
Intracardiac mass (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 3 | 1 | 2 | 0 | 0 | 3 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 2 | 7 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chalazion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chorioretinopathy (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 3 | 2 | 0 | 2 | 2 | 2
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Keratopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation decreased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 2 | 3 | 2 | 5 | 5 | 10 | 5 | 4 | 3 | 4 | 6 | 5
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1 | 5 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 5 | 0 | 3 | 3 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 1 | 3 | 3 | 2 | 2 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 4 | 1 | 15 | 6 | 11 | 12 | 4 | 5 | 5 | 10 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 7 | 4 | 4 | 10 | 1 | 1 | 0 | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 9 | 6 | 26 | 6 | 15 | 15 | 7 | 1 | 6 | 11 | 7
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 9 | 8 | 32 | 15 | 18 | 27 | 10 | 5 | 6 | 18 | 12
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 9 | 3 | 8 | 7 | 6 | 0 | 2 | 6 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 4 | 5 | 3 | 7 | 7 | 2 | 1 | 0 | 6 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 4 | 3 | 0 | 1 | 1 | 1 | 1 | 1 | 3
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 6 | 1 | 4 | 4 | 0 | 1 | 0 | 0 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 2 | 11 | 12 | 49 | 11 | 30 | 26 | 11 | 5 | 10 | 26 | 21
Oral mucosa erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 2 | 2
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 4 | 2 | 6 | 12 | 39 | 8 | 23 | 26 | 13 | 3 | 8 | 20 | 21
Asthenia (General disorders) | 0 | 0 | 8 | 3 | 12 | 3 | 2 | 6 | 1 | 1 | 0 | 6 | 3
Axillary pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Chills (General disorders) | 3 | 3 | 9 | 11 | 38 | 8 | 24 | 29 | 6 | 2 | 5 | 15 | 13
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Fatigue (General disorders) | 5 | 4 | 13 | 12 | 50 | 22 | 35 | 32 | 12 | 7 | 4 | 29 | 16
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 1
Influenza like illness (General disorders) | 0 | 0 | 3 | 2 | 3 | 4 | 12 | 6 | 5 | 2 | 3 | 3 | 6
Malaise (General disorders) | 0 | 0 | 0 | 2 | 7 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 1
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 4 | 2 | 0 | 3 | 2 | 0 | 0 | 0 | 1 | 1
Nodule (General disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2 | 3 | 2 | 2 | 3 | 1 | 0 | 1 | 0 | 2
Oedema peripheral (General disorders) | 1 | 0 | 6 | 5 | 18 | 9 | 13 | 14 | 7 | 3 | 2 | 10 | 11
Pain (General disorders) | 2 | 2 | 4 | 4 | 8 | 4 | 6 | 4 | 0 | 2 | 0 | 3 | 3
Peripheral swelling (General disorders) | 0 | 0 | 1 | 1 | 4 | 1 | 4 | 3 | 1 | 1 | 2 | 1 | 1
Pyrexia (General disorders) | 3 | 4 | 10 | 13 | 58 | 13 | 39 | 37 | 12 | 7 | 7 | 19 | 19
Swelling (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 2 | 2 | 1 | 2 | 3 | 2 | 1 | 0 | 1 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 4 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 4 | 1 | 1 | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 2 | 3 | 1 | 3 | 4 | 3 | 1 | 0 | 4 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 3 | 3 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 1 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1 | 4 | 0 | 3 | 5 | 0 | 1 | 3 | 5 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 5 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1
Periorbital infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1
Rash pustular (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 5 | 7 | 0 | 2 | 4 | 1 | 0 | 0 | 3 | 6
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 10 | 5 | 10 | 5 | 5 | 2 | 3 | 4 | 6
Urinary tract infection (Infections and infestations) | 1 | 0 | 5 | 4 | 18 | 3 | 3 | 8 | 6 | 2 | 2 | 5 | 10
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 3 | 1 | 0 | 1 | 0 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 3 | 0 | 3 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 2 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 3 | 7 | 1 | 11 | 6 | 2 | 1 | 3 | 8 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 4 | 12 | 1 | 10 | 10 | 3 | 0 | 3 | 6 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 2 | 14 | 2 | 11 | 7 | 2 | 0 | 5 | 5 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 5 | 2 | 4 | 1 | 1 | 1 | 0 | 4 | 5
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Carbon dioxide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 1 | 6 | 0 | 1 | 5 | 1 | 0 | 1 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 3 | 3 | 12 | 1 | 11 | 6 | 6 | 0 | 3 | 6 | 6
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 0 | 2 | 1 | 5 | 2 | 1 | 0 | 0 | 2 | 2
Mean cell volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 2 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 2 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 3
Protein urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroxine free decreased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 0 | 2 | 1 | 1
Weight decreased (Investigations) | 0 | 0 | 3 | 0 | 5 | 4 | 8 | 6 | 3 | 1 | 2 | 4 | 3
Weight increased (Investigations) | 0 | 1 | 5 | 2 | 3 | 0 | 1 | 4 | 2 | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 2 | 7 | 23 | 11 | 18 | 16 | 7 | 2 | 3 | 12 | 14
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3 | 2 | 12 | 1 | 4 | 5 | 2 | 1 | 1 | 5 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 8 | 3 | 6 | 5 | 0 | 0 | 1 | 4 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 4 | 4 | 0 | 2 | 0 | 0 | 2 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 6 | 1 | 4 | 3 | 1 | 0 | 2 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 13 | 3 | 1 | 5 | 1 | 1 | 3 | 5 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 7 | 1 | 1 | 3 | 1 | 0 | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 11 | 1 | 5 | 7 | 1 | 0 | 2 | 5 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 8 | 4 | 5 | 2 | 1 | 0 | 0 | 6 | 2
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 6 | 6 | 18 | 18 | 28 | 19 | 12 | 9 | 8 | 17 | 17
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 6 | 13 | 6 | 7 | 12 | 8 | 1 | 4 | 4 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 7 | 2 | 0 | 3 | 0 | 0 | 3 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 5 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5 | 2 | 13 | 2 | 3 | 11 | 2 | 1 | 0 | 7 | 5
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 3 | 6 | 0 | 7 | 7 | 4 | 1 | 2 | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 3 | 1 | 3 | 2 | 2 | 0 | 0 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 8 | 6 | 4 | 6 | 0 | 1 | 1 | 4 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 6 | 17 | 12 | 16 | 12 | 2 | 1 | 3 | 12 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 5 | 5 | 4 | 7 | 2 | 2 | 0 | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 5 | 16 | 11 | 11 | 13 | 5 | 4 | 2 | 5 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 3 | 5 | 3 | 5 | 0 | 3 | 3 | 1 | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 1 | 3 | 0 | 3 | 7 | 0 | 2 | 0 | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1 | 3 | 4 | 5 | 0 | 1 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2 | 4 | 5 | 7 | 6 | 0 | 4 | 1 | 4 | 6
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1 | 2 | 2 | 8 | 4 | 2 | 0 | 1 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 4 | 5 | 24 | 5 | 12 | 10 | 7 | 4 | 1 | 14 | 4
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 5 | 0 | 5 | 5 | 1 | 1 | 1 | 2 | 3
Dyskinesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 3 | 12 | 8 | 32 | 17 | 25 | 18 | 9 | 5 | 4 | 13 | 16
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1 | 1 | 4 | 1 | 3 | 4 | 1 | 2 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 1 | 2 | 0 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 5 | 0 | 2 | 1 | 2 | 0 | 1 | 2 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 3 | 1 | 6 | 4 | 4 | 4 | 1 | 2 | 0 | 1 | 0
Noninfective encephalitis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 6 | 6 | 0 | 4 | 3 | 2 | 1 | 1 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 1 | 1 | 1 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 3 | 1 | 3 | 3 | 1 | 0 | 1 | 4 | 3
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 5 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 5 | 1 | 10 | 5 | 5 | 4 | 2 | 0 | 2 | 0 | 2
Confusional state (Psychiatric disorders) | 1 | 1 | 2 | 0 | 5 | 1 | 3 | 6 | 1 | 0 | 1 | 4 | 2
Depression (Psychiatric disorders) | 0 | 0 | 1 | 4 | 6 | 2 | 5 | 4 | 1 | 0 | 1 | 2 | 3
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 6 | 6 | 4 | 7 | 10 | 0 | 2 | 2 | 3 | 4
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 4 | 0 | 1 | 4 | 0 | 0 | 1 | 2 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 1 | 4
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 1 | 0 | 1 | 0 | 3 | 2
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5 | 9 | 22 | 11 | 10 | 19 | 5 | 5 | 4 | 14 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 1 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 3 | 12 | 4 | 7 | 7 | 5 | 1 | 2 | 5 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 5 | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 6 | 0 | 2 | 5 | 1 | 1 | 1 | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 7 | 1 | 6 | 6 | 2 | 1 | 1 | 4 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 1 | 16 | 0 | 7 | 9 | 3 | 1 | 2 | 3 | 5
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 9 | 3 | 1 | 2 | 1 | 2 | 4
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 4 | 4 | 1 | 1 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 4 | 2 | 1 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 2 | 0 | 1 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 4 | 0 | 3 | 2 | 1 | 2 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 3 | 11 | 6 | 6 | 12 | 1 | 0 | 2 | 4 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 8 | 19 | 8 | 3 | 5 | 4 | 4 | 5 | 2
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 5 | 12 | 2 | 6 | 10 | 0 | 3 | 4 | 6 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 2 | 5 | 2 | 6 | 11 | 3 | 3 | 1 | 6 | 6
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 1 | 3 | 0 | 2 | 4 | 2 | 2 | 1 | 1 | 2
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 7 | 5 | 1 | 5 | 10 | 2 | 1 | 1 | 1 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 3 | 1 | 3 | 0 | 2 | 2
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 3 | 1 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 1 | 10 | 1 | 5 | 6 | 1 | 2 | 0 | 6 | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 4 | 15 | 5 | 9 | 1 | 3 | 2 | 4 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 7 | 16 | 3 | 11 | 15 | 3 | 1 | 3 | 8 | 9
Nodular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3 | 9 | 4 | 4 | 2 | 0 | 2 | 2 | 3
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 5 | 1 | 2 | 2 | 0 | 1 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 3 | 3 | 2 | 1 | 0 | 0 | 2 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 1 | 4 | 8 | 8 | 8 | 3 | 3 | 2 | 4 | 7
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 4 | 4 | 7 | 4 | 2 | 4 | 2 | 4 | 6 | 4
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 6 | 9 | 21 | 19 | 13 | 18 | 8 | 4 | 6 | 14 | 18
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1 | 1 | 0 | 5 | 1 | 2 | 1 | 1 | 2 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 2 | 4 | 0 | 5 | 3 | 2 | 6 | 1 | 1 | 0 | 1 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 3 | 2 | 2 | 5 | 2 | 0 | 4 | 0 | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 5 | 3 | 5 | 4 | 2 | 3 | 1 | 5 | 7
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 1 | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 4 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 5 | 1 | 2 | 1 | 0 | 1 | 2 | 2 | 4
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Flushing (Vascular disorders) | 1 | 0 | 1 | 0 | 7 | 4 | 6 | 1 | 1 | 0 | 1 | 1 | 4
Hot flush (Vascular disorders) | 1 | 0 | 2 | 0 | 2 | 1 | 5 | 4 | 0 | 2 | 0 | 1 | 5
Hypertension (Vascular disorders) | 0 | 0 | 2 | 3 | 6 | 2 | 4 | 9 | 4 | 0 | 0 | 7 | 7
Hypotension (Vascular disorders) | 1 | 1 | 3 | 2 | 9 | 0 | 2 | 4 | 0 | 2 | 0 | 3 | 5
Labile blood pressure (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 4 | 1 | 1 | 2 | 2 | 3
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.